

# CM4620-205 Protocol

# A Single-Blind Dose-Ranging Pharmacodynamic Study of Auxora for the Treatment of Patients with Critical COVID-19 Pneumonia

Version: 3.1

Issue Date: November 18, 2021

Clinical Trial Number: NCT04661540



# CM4620-205

# A Single-Blind Dose-Ranging Pharmacodynamic Study of Auxora for the Treatment of Patients with Critical COVID-19 Pneumonia

**Sponsor**: CalciMedica, Inc.

505 Coast Boulevard South, Suite 307

La Jolla, CA 92037

Sponsor Medical Contact: Sudarshan Hebbar, MD

(816) 838-7105 – Mobile

sudarshan@calcimedica.com – Email

#### FOR QUALIFIED INVESTIGATORS AND THEIR IRB/EC ONLY

Version: 3.1

Issue Date: November 18, 2021

#### **Confidentiality Statement**

The information contained in this document is confidential and proprietary property of CalciMedica, Inc. Any distribution, copying, or disclosure is strictly prohibited unless federal regulations or state law requires such disclosure. Prior written authorization of CalciMedica, Inc. is required for any disclosure or use of the information contained herein. Persons to whom the information is disclosed must know that it is confidential and that it may not be further disclosed by them.

# SPONSOR APPROVAL AND SIGNATURE PAGE

| Som When | 01-December-2021 |
|------------------------------------------------------|------------------|
| Sudarshan Hebbar MD<br>Chief Medical Officer | Date |
| Zumeth A. Handerman | 01-December-2021 |
| Kenneth A. Stauderman Ph.D. Chief Scientific Officer | Date |

# **SYNOPSIS**

| <b>Protocol Number:</b> | CM4620-205 | | |
|---|---|---|---|
| Protocol Title for Part 2: | A Single-Blind Dose-Ranging Pharmacodynamic Study of Auxora for the Treatment of Patients with Critical COVID-19 Pneumonia | | |
| Sponsor: | CalciMedica, Inc.<br>505 Coast Blvd. South, Suite 307<br>La Jolla, CA 92037 USA | | |
| <b>Study Phase:</b> | 2 | | |
| Number of Patients and Sites: | | atients with confirmed COVID-<br>l ventilation randomized at up to | - |
| Study Drug Dose | Cohort | Auxora | Placebo |
| and Route of Administration: | 1 | Day 1: 1.25 mL/kg<br>Day 2: 1.0 mL/kg<br>Day 3: 1.0 mL/kg | Day 1: 1.25 mL/kg<br>Day 2: 1.0 mL/kg<br>Day 3: 1.0 mL/kg |
| | Day 1: 1.25 mL/kg Day 2: 1.25 mL/kg Day 2: 1.25 mL/kg Day 3: 1.0 mL/kg Day 3: 1.0 mL/kg Day 4: 1.0 mL/kg Day 4: 1.0 mL/kg | | |
| | 3 | Day 1: Initial infusion of<br>1.25 mL/kg over 4 hours<br>After initial infusion completed,<br>start continuous infusion of<br>1.0 mL/kg up to 24 hours for 96<br>hours | |
| | 0 hours. Ir (±2) and 4 administer be adminis | Start of the First Infusion of Study Drug (SFISD) will be considered ars. In Cohorts 1 and 2, study drug will again be administered at 24 and 48 (±2) hours from the SFISD. In Cohort 2 study drug will also be nistered at 72 (±2) hours from the SFISD. In Cohort 3, study drug will ministered as a continuous infusion for 96 hours after the first infusion drug drug is completed. Shorts 1, 2, and for the first infusion in Cohort 3, study drug will be nistered intravenously as a continuous infusion over 4 hours (± 30 tes). In Cohort 3, after the end of the first infusion, a 96-hour nuous infusion will commence; during the continuous infusion study infusion bags will be prepared daily, each diluted up to 500 mL with didition of normal saline and each for administration continuously up to burs (± 30 minutes). Study drug will be administered via a bag and g compatible with lipid emulsions and using a 1.2-micron filter. | |
| | administer<br>minutes). I<br>continuous<br>drug infus<br>the addition<br>24 hours (s | | |
| | | The SFISD should occur within 12 hours of the patient or LAR providing informed consent. The dosing will be based on actual body weight obtained | |

at the time of hospitalization or screening for the study, whichever is the most recent weight at randomization.

As described in the pharmacy manual, there will be an upper limit of the absolute dose (volume) of Auxora and volume of Placebo that will be administered for patients weighing more than 125kg. The concentration of CM4620 in Auxora is 1.6 mg/kg.

### **Hypothesis:**

Recently published results suggest SARS-CoV-2 causes a slowly unfolding, spatially-limited alveolitis in which alveolar macrophages harboring SARS-CoV-2 transcripts and T cells producing IFN- $\gamma$  form a positive feedback loop that drives progressive alveolar inflammation. T cell activation and the production of IFN- $\gamma$ , as well as other pro-inflammatory cytokines such as IL-6, IL-17, and TNF $\alpha$ , are mediated via calcium entry through calcium release-activated calcium (CRAC) channels.

Auxora is a calcium release-activated calcium (CRAC) channel inhibitor that potently blocks the production and release of pro-inflammatory cytokines from immune cells and may further directly protect the lung through a local effect on CRAC channels and modulation of NFAT-induced activation of the lung endothelium. In vivo efficacy data shows that treatment with Auxora decreases the levels of lung IL-6, TNF $\alpha$ , and myeloperoxidase (MPO) mRNA production in animals with experimental acute pancreatitis, a common cause of ARDS. In a Phase 2a study of patients with acute pancreatitis and accompanying SIRS with hypoxemia at presentation, treatment with Auxora resulted in a significant reduction in elevated serum IL-6 levels and improved oxygenation. Data from the open-label Part 1 of a Phase 2a study showed improved outcomes and decreased need for mechanical ventilation in patients treated with Auxora who had severe Covid-19 pneumonia and were receiving low flow supplemental oxygen.

Auxora is given intravenously, is distributed into the lung within 2 to 4 hours of the start of infusion, has a rapid onset of activity with stimulated IL-2 release being decreased by >50% at the end of the infusion, and does not appear to have long term immune-modulatory effects with recovery of IL-2 release 24-48 hours after the end of the infusion.

Auxora holds promise as a potential treatment for patients with critical COVID-19 pneumonia and Auxora may also prove to a beneficial treatment in other forms of ARDS. Further studies to define the optimal dose for patients with ARDS are needed.

| <b>Objectives:</b> | Primary: |
|---|---|
| ~ <b>,</b> | To assess the pharmacodynamic response of bronchoalveolar lavage (BAL) T cell/monocyte subsets and chemokine release to various doses of Auxora in patients with critical COVID-19 pneumonia |
| | Secondary: |
| | <ul> <li>To assess the safety and tolerability of Auxora in patients with critical<br/>COVID-19 pneumonia</li> </ul> |
| | • To assess the serum and BAL pharmacokinetic profile of various doses of Auxora in patients with critical Covid-19 pneumonia |
| Inclusion Criteria: | All of the following must be met for a patient to be randomized into the study: |
| | 1. Has laboratory-confirmed SARS-CoV-2 infection as determined by polymerase chain reaction (PCR) or other commercial or public health assay in any specimen; |
| | 2. Moderate ARDS characterized by the following criteria: |
| | <ul> <li>Invasive mechanical ventilation with a minimum PEEP of 5 cm<br/>H<sub>2</sub>O;</li> </ul> |
| | <ul> <li>PaO<sub>2</sub>/FiO<sub>2</sub> ≤200 that may be estimated from pulse oximetry or<br/>determined by arterial blood gas;</li> </ul> |
| | <ul> <li>No evidence of volume overload or heart failure as the sole cause of<br/>pulmonary edema;</li> </ul> |
| | 3. The patient is $\geq$ 18 years of age at the time of consent; |
| | 4. QTcF interval ≤ 440 milliseconds; |
| | 5. A female patient of childbearing potential must not attempt to become pregnant for 39 months, and if sexually active with a male partner, is willing to practice acceptable methods of birth control for 39 months after the last dose of study drug; |
| | 6. A male patient who is sexually active with a female partner of childbearing potential is willing to practice acceptable methods of birth |

must not donate sperm for 39 months;

control for 39 months after the last dose of study drug. A male patient

representative (LAR) who is willing and able to, provide informed consent to participate, and to cooperate with all aspects of the protocol.

7. The patient is willing and able to, or has a legal authorized

### **Exclusion Criteria:**

Patients with any of the following conditions or characteristics must be excluded from randomizing:

- 1. Expected survival or time to withdrawal of life-sustaining treatments expected to be <7 days.
- 2. ECMO;
- 3. Invasive mechanical ventilation for more than 7 days
- 4. Suspected septic shock;
- 5. The patient has a history of:
  - a. Organ or hematologic transplant;
  - b. HIV;
  - c. Active hepatitis B or hepatitis C infection;
- 6. Current treatment with:
  - a. Chemotherapy;
  - b. Immunosuppressive medications or immunotherapy (see Section 5.3 for list of prohibited immunosuppressive medications and immunotherapy) at the time of consent;
  - c. Hemodialysis or Peritoneal Dialysis;
- 7. The patient is known to be pregnant or is nursing;
- 8. Currently participating in another study of an investigational drug or therapeutic medical device at the time of consent;
- 9. Allergy to eggs or any of the excipients in study drug.

#### **Study Design:**

This will be a single-blind study where the patient will not know if they are receiving Auxora or Placebo. The first 4 patients will be enrolled in Cohort 1 and randomized 3:1 to Auxora or Placebo. If dose escalation occurs, the next 4 patients will be enrolled in Cohort 2 and randomized 3:1 to Auxora or Placebo. If dose escalation continues, the next 8 patients will be enrolled in Cohort 3 and randomized 3:1 to Auxora or Placebo. The decision to escalate dosing will be made by CalciMedica in consultation with the PI after the review of safety events in Cohorts 1 and 2.

Consultation between the PI and CalciMedica will occur if any patient receiving Auxora in Cohorts 1, 2 or 3 experiences one of the cardiac conduction events listed below during the 144 hours after the Start of the First Infusion of Study Drug (SFISD):

- OTcF interval of > 500 msec; or
- QTcF prolongation of  $\geq$  60 msec as compared to baseline; or
- Mobitz Type II second degree atrioventricular (AV) block; or

- Third degree or high grade AV block; or
- Polymorphic Ventricular Tachycardia;

If one of the listed safety events occurs in a patient who is receiving Auxora in Cohort 1 but the event is not thought to be dose limiting, 4 additional patients will be enrolled in Cohort 1 and randomized 3:1 to Auxora versus Placebo for a total of 8 patients enrolled in the cohort, 6 randomized to Auxora and 2 to Placebo. The PI and CalciMedica will consult after all 8 patients are enrolled to determine if dose escalation to Cohort 2 will occur. If one of the listed safety events occurs in a patient who is receiving Auxora in Cohort 1 and the event is dose limiting, further dosing will not occur using the planned dose regimens but may occur using a regimen that provides lower total exposure of drug.

If one of the listed safety events occurs in a patient who is receiving Auxora in Cohort 2 but the event is not thought to be dose limiting, 4 additional patients will be enrolled in Cohort 2 and randomized 3:1 to Auxora versus Placebo for a total of 8 patients enrolled in the cohort, 6 randomized to Auxora and 2 to Placebo. The PI and CalciMedica will consult after all 8 patients are enrolled to determine if dose escalation to Cohort 3 will occur. If one of the listed safety events occurs in a patient who is receiving Auxora in Cohort 2 and the event is dose limiting, further dosing will not occur in either Cohorts 2 or 3. 4 additional patients may be enrolled in Cohort 1 and randomized 3:1 to Auxora versus Placebo. The 4 additional patients in Cohort 1 will receive a dose regimen of an initial infusion followed by continuous infusion for 48 hours.

If one of the listed safety events occurs in a patient who is receiving Auxora in Cohort 3 but the event is not felt to be dose limiting, 4 additional patients will be enrolled in Cohort 3 and randomized 3:1 to Auxora versus Placebo for a total of 12 patients enrolled in the cohort, 9 randomized to Auxora and 3 to Placebo. If one of the listed safety events occurs in a patient who is receiving Auxora in Cohort 3 and the event is dose limiting, further dosing will not occur in Cohort 3. 4 additional patients may be enrolled in Cohort 2 and randomized 3:1 to Auxora versus Placebo. The 4 additional patients in Cohort 2 will receive a dose regimen of an initial infusion followed by continuous infusion for 72 hours.

A study physician or appropriately trained delegate will perform assessments at Screening, immediately prior to the SFISD, and then every 24 hours (±1 hours) until 240 hours after the SFISD. After 240 hours from the SFISD, the patient will be assessed q48 hours until Day 30 after the SFISD, or until discharge if earlier. Patients who are discharged before Day 25 after the SFISD will be followed-up at Day 30 (±5 days). Patients will be followed up at Day 60 (±5 days). for a safety and mortality assessment.

This assessment will be conducted by phone for patients discharged prior to Day 55.

Fluid from a bronchoalveolar lavage (BAL) should be obtained prior to the SFISD (-12 hours) and then again 24 (±12) hours after the last infusion of study drug in Cohorts 1 and 2. In Cohort 3, BAL fluid will be obtained during the final 24 hours of the continuous infusion. BAL fluid will be used for flow cytometry, single cell RNA sequencing, and chemokine/biomarker panel. On the BAL fluid obtained from the second BAL, CM4620 levels will be determined in patients receiving Auxora.

ECGs will be performed and QTcF will recorded daily at each assessment until 144 (+2) hours from the SFISD. If at any time QT prolongation is suspected on a cardiac monitor, a ECG will be performed and QTcF will be recorded. Blood specimen for PK analysis should be obtained in patients receiving Auxora.

All patients enrolled in the study should receive care consistent with local standard of care including for ventilator management. Patients should receive conservative intravenous fluid strategies such as FACTT LITE. All patients should receive pharmacological prophylaxis to prevent the development of venous thromboembolic disease. The type and dose of prophylaxis should be determined by local standard of care.

Patients enrolled in the study should receive dexamethasone as standard of care. If patients are not receiving dexamethasone at the time of randomization, starting dexamethasone during the hospitalization should be considered. If the patient is already receiving dexamethasone at the time of randomization, dexamethasone should be continued on its established dosing schedule. The COVID-19 Treatment Guidelines Panel of the National Institutes of Health recommends using dexamethasone (at a dose of 6 mg per day, given orally or intravenously, for up to 10 days) in patients with COVID-19 who require supplemental oxygen. Before initiating dexamethasone, the potential risks and benefits of administering corticosteroids should be assessed including risks for hyperglycemia and secondary infections. At this time, it is not known whether other corticosteroids, such as prednisone, methylprednisolone, or hydrocortisone, will have a similar benefit to dexamethasone. Of note, the dose equivalencies for dexamethasone 6 mg daily are prednisone 40 mg, methylprednisolone 32 mg, and hydrocortisone 160 mg.

If patients are not receiving remdesivir at the time of randomization, starting remdesivir during the hospitalization may be considered. If the patient is already receiving remdesivir at the time of randomization, remdesivir should be continued on its established dosing schedule. The suggested dose of remdesivir for adults weighing ≥40 kg and not requiring invasive

mechanical ventilation and/or ECMO is a single dose of 200 mg infused intravenously over 30 to 120 minutes on Day 1 followed by once-daily maintenance doses of 100 mg infused intravenously over 30 to 120 minutes for 4 days (days 2 through 5). If a patient does not demonstrate clinical improvement, treatment may be extended for up to 5 additional days (i.e., up to a total of 10 days). Auxora and remdesivir should not be infused at the same time but should be given sequentially.

Patients may also be considered for the administration of convalescent plasma in the study as per local standard of care.

Immunosuppressive medications or immunotherapies are prohibited in patients randomized into the study (see Section 5.3 for a list of prohibited medication). The use of dextromethorphan in patients is discouraged when enrolled in the study.

### Pharmacodynamic Assessments

- Blood biomarkers and chemokines;
- On fluid collected from the BAL performed prior to the SFISD (-12 hours) and 24 (±12) hours after completing the last infusion of study drug in Cohorts 1 and 2 and during the final 24 hours of the continuous infusion in Cohort 3:
  - o Flow cytometry
  - o Single cell RNA sequencing
  - o Biomarker/Chemokine Panel
  - o SARS-CoV-2 PCR with semiguantitation (cT value)

# Pharmacokinetic Assessments:

- Plasma levels of CM4620 obtained from blood samples at selected timepoints in patients receiving Auxora
- Level of CM4620 in fluid collected from the BAL performed 24 (±12) hours after the last infusion of study drug in Cohorts 1 and 2 and during the final 24 hours of the continuous infusion in Cohort 3

# Pharmacodynamic Endpoint:

- Proportion of immune cells in BAL fluid (specifically: Tregs, CD4 and CD8 T cells, B cells, NK cells, alveolar macrophages monocytes, and neutrophils). T cell activation will also be assessed via flow cytometry by assessing surface expression of HLA-DR and CD127.
- Activation of all immune cell types will be assessed using integrative analysis of single cell RNA sequencing on all subjects across all time points. After demultiplexing reads will be aligned to a hybrid genome containing human (GRCh38) and SARS-CoV-2 (NC\_045512.2) reference genomes. Resulting cell-by-gene matrices from all samples will be normalized using sctransform algorithm and integrated using BBKNN or scVI/scANVI approach followed by Leiden clustering, identification of marker genes for each cluster and assigning cell type identity to clusters (for details see Grant et al., 2021). It will be assessed whether treatment with Auxora resulted in emergence of the new

| | clusters/cell types/cell states and markers characterizing these newly emergent populations will be evaluated. For homologous cell types differential genes expression analysis will be performed between Auxora- and placebo-treated subjects, split by time-points. The impact of Auxora treatment on detection of SARS-CoV-2 positive and negative strand RNA in infected cells will also be assessed. Differential gene expression will be performed on per-cluster level and using multilevel statistics (per-cluster and per subject level, to assess biological variability within the group). |
|---|---|
| Efficacy Endpoints: | <ul> <li>All-Cause Mortality at Day 60</li> <li>Number of Days on Mechanical Ventilation after randomization</li> <li>Number of Days in the Hospital after randomization</li> <li>Number of Days in the ICU after randomization</li> </ul> |
| Safety Endpoints: | <ul> <li>Pre-defined changes in cardiac conduction</li> <li>The incidence of TEAEs and SAEs</li> <li>The intensity and relationship of TEAEs and SAEs</li> <li>Mortality at Day 30</li> </ul> |
| Sample Size<br>Calculation: | Sample size considerations were based on precision estimates and the ability to construct 95% confidence intervals around point estimates for pharmacodynamics endpoints with reasonable precision. Sample sizes as small as 9 patients per arm will allow for construction of 95% confidence intervals with half-widths as small as 0.77 standard deviation units. For other assessments, the study is not powered for analysis with inferential statistics. All data will be summarized using descriptive statistics only. Continuous data will be summarized with number of patients (n), mean, median, minimum, maximum, standard of deviation, coefficient of variation and or geometric mean. Categorical data will be summarized with number and proportion of patients. |

# **Table of Contents**

| Spo | onsor A | Approval and Signature Page | 2 |
|---|---|---|---|
| Syı | nopsis | | 3 |
| Lis | t of Ta | ıbles | 14 |
| Lis | t of Te | erms and Abbreviations | 15 |
| 1 | INTE | RODUCTION | 17 |
| | 1.1 | COVID-19 | 17 |
| | 1.2 | Overview of CM4620 | 18 |
| | 1.3 | Pre-Clinical Development of CM4620 | 18 |
| | | 1.3.1 Pre-Clinical Safety and Toxicology Studies | 18 |
| | | 1.3.2 Preclinical Efficacy Studies | 19 |
| | 1.4 | Clinical Development of Auxora | 19 |
| | | 1.4.1 Single Ascending Dose and Multiple Ascending Dose Studies | 19 |
| | | 1.4.2 Open Label Study in Patients with Acute Pancreatitis with Accompanying SIRS and Hypoxemia (CM4620-201) | |
| | 1.5 | Pharmacodynamic and Pharmacokinetic Study in Patients with Acute Pancreatitis (CM4620-202) | |
| | 1.6 | Study in Severe Covid-19 Pneumonia (CM4620-204) | 24 |
| | 1.7 | Rationale for Current Study and Selected Doses | 25 |
| 2 | OBJI | ECTIVES AND ENDPOINTS | 26 |
| | 2.1 | Primary Objective | 26 |
| | 2.2 | Secondary Objectives | 26 |
| | 2.3 | Endpoints | 26 |
| 3 | INVI | ESTIGATIONAL PLAN | 27 |
| | 3.1 | Study Design | 27 |
| | 3.2 | End of Study | 28 |
| | 3.3 | Sponsor Termination of the Study | 28 |
| 4 | SELI | ECTION OF PATIENTS | 29 |
| | 4.1 | Inclusion Criteria | 29 |
| | 4.2 | Exclusion Criteria | 29 |
| | 4.3 | Re-Screening. | 30 |
| 5 | TRE | ATMENT OF PATIENTS | 31 |
| | 5.1 | Overview | 31 |
| | 5.2 | Discharge Criteria | 31 |
| | 5.3 | Prohibited Medications | 32 |

| | 5.4 | Compliance | 32 |
|---|------|------------------------------------------------------|----|
| 6 | PRO | CEDURES | 33 |
| | 6.1 | Enrollment Procedures | 33 |
| | 6.2 | Discontinuation and Withdrawal | 33 |
| 7 | STUI | DY DRUG MATERIALS AND MANAGEMENT | 34 |
| | 7.1 | Auxora Product Description | 34 |
| | 7.2 | Placebo Product Description | 34 |
| | 7.3 | Auxora and Placebo Storage | 34 |
| | 7.4 | Auxora and Placebo Preparation | 34 |
| | 7.5 | Auxora and Placebo Administration | 35 |
| | 7.6 | Packaging and Labeling | 35 |
| | 7.7 | Accountability, Handling and Disposal | 36 |
| 8 | VISI | TS AND STUDY SPECIFIC ASSESSMENTS | 37 |
| | 8.1 | Screening | 37 |
| | 8.2 | Baseline Assessment | 37 |
| | 8.3 | Randomization | 37 |
| | 8.4 | Start of First Infusion of Study Drug (SFISD) 0 hour | 37 |
| | 8.5 | 24 hours | 38 |
| | 8.6 | 48 hours | 38 |
| | 8.7 | 72 hours | 39 |
| | 8.8 | 96 hours | 39 |
| | 8.9 | 120 hours | 40 |
| | 8.10 | 144 hours | 40 |
| | 8.11 | 168 hours Until Discharge or Day 30 if Earlier | 41 |
| | 8.12 | Day 60 and Day 30 | 41 |
| | 8.13 | Study Assessments | 41 |
| | | 8.13.1 Concomitant Medications | 41 |
| | | 8.13.2 Vital Signs | 41 |
| | | 8.13.3 PO <sub>2</sub> /FiO <sub>2</sub> | 41 |
| | | 8.13.4 Laboratory Analyses | 42 |
| | | 8.13.5 PK Samples | 42 |
| | | 8.13.6 Blood Biomarkers and Chemokines | 42 |
| | | 8.13.7 BAL Fluid | 43 |
| | | 8.13.8 Nasopharyngeal SARS-CoV-2 PCR | 43 |

| 9 | ADV | ERSE EVENTS | 44 |
|---|---|---|---|
| | 9.1 | Definition of Adverse Event | 44 |
| | 9.2 | Definition of Serious Adverse Event | 44 |
| | 9.3 | Eliciting Adverse Event Information | 45 |
| | 9.4 | Recording Adverse Events | 45 |
| | 9.5 | Assessment of Relationship to Study Drug | 46 |
| | 9.6 | Assessment of Severity | 46 |
| | 9.7 | Reporting of Serious Adverse Events | 46 |
| | 9.8 | Suspected Pregnancy in a Woman of Childbearing Potential | 48 |
| 10 | STAT | TISTICAL METHODS | 50 |
| | 10.1 | General Considerations | 50 |
| | 10.2 | Study Endpoints | 50 |
| | 10.3 | Analysis Sets | 51 |
| | | 10.3.1 Pharmacodynamic and Efficacy Analysis Set | 51 |
| | | 10.3.2 Safety Analysis Set | 51 |
| | 10.4 | Disposition | 51 |
| | 10.5 | Analysis of Demographic and Baseline Data | 51 |
| | 10.6 | PD Analysis | 51 |
| | | 10.6.1 Mortality at Day 60 and Day 30 | 52 |
| | | 10.6.2 Number of Days in the Hospital | 52 |
| | | 10.6.3 Number of Days in the ICU and Days on Mechanical Ventilation | 52 |
| | 10.7 | Safety Analysis | 52 |
| | 10.8 | PK Analysis | 53 |
| 11 | ADM | INISTRATIVE CONSIDERATIONS | 54 |
| | 11.1 | Monitoring of the Study | 54 |
| | 11.2 | Inspection of Records | 54 |
| | 11.3 | Study Record Retention | 54 |
| | 11.4 | Study Conduct: Good Clinical Practice and Declaration of Helsinki | 54 |
| | 11.5 | Responsibilities of the Investigator and the IRB/EC | 54 |
| | 11.6 | Confidentiality | 55 |
| | 11.7 | Modification of the Protocol. | 55 |
| | 11.8 | Informed Consent. | 56 |
| | 11.9 | Protocol Violations and Deviations | 56 |
| | 11.10 | Financial Disclosure. | 57 |
| | 11.11 | Sponsor Obligations | 57 |

| 11.12 Investigator Documentation | 57 |
|---|---|
| 11.13 Clinical Study Insurance | 57 |
| 11.14 Use of Information | 58 |
| 11.15 Publications | 58 |
| 11.16 Independent Data Monitoring Committee | 58 |
| 12 REFERENCES | 59 |
| Appendix 1. Imputed PaO <sub>2</sub> /FiO <sub>2</sub> Ratio | 60 |
| Appendix 2. Schedule of Events | 61 |
| List of Tables | |
| Table 1. SAD (CM4620-101) | 19 |
| Table 2. MAD (CM4620-102) | |
| Table 3. Demographics and Baseline Characteristics of Patients in CM4620-201 | 23 |
| Table 4. Auxora Product Information | 34 |
| Table 5 Conversion of O2 Flow to FiO2 | 42. |

PK

# **List of Terms and Abbreviations**

| Abbreviation | Definition |
|---|---|
| AE | adverse event |
| ALT | alanine transaminase |
| AP | acute pancreatitis |
| ARDS | acute respiratory distress syndrome |
| AST | aspartate transaminase |
| BAL | bronchoalveolar lavage |
| CFR | Code of Federal Regulations |
| COVID-19 | Disease from infection with coronavirus 2019 or SARS-CoV-2 |
| CPK | creatine kinase |
| CRAC | calcium release-activated calcium |
| CRF | case report form |
| ECG | electrocardiogram |
| ECMO | Extracorporeal Membrane Oxygenation |
| EDTA | edetate disodium salt dehydrate |
| FAEE | fatty acid ethyl ester |
| FiO <sub>2</sub> | fraction of inspired oxygen |
| GMP | Good Manufacturing Practice of Medicinal Products |
| Hr(s) | hour(s) |
| ICH | International Conference on Harmonization |
| IDMC | Independent Data Monitoring Committee |
| IRB | Institutional Review Board |
| IV | intravenous |
| Kg | kilogram |
| L | liter |
| LAR | legal authorized representative |
| LDH | lactate dehydrogenase |
| LTVV | low tidal volume ventilation |
| MAD | multiple ascending dose |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MPO | myeloperoxidase |
| NOAEL | no observable adverse effect level |
| PaO <sub>2</sub> | Partial Pressure of Oxygen (arterial) |
| PCR | polymerase chain reaction |
| PI | Principal Investigator |

pharmacokinetic

| Abbreviation | Definition |
|--------------|-------------------------------------------------|
| PT | preferred Term |
| QTcF | QT corrected for HR using Fridericia's method |
| SAD | single ascending dose |
| SAE | Serious adverse event |
| SARS | severe acute respiratory syndrome |
| SARS-CoV-2 | severe acute respiratory syndrome coronavirus 2 |
| SC | Supportive Care |
| SFISD | Start of First Infusion of Study Drug |
| SIRS | Systemic inflammatory response syndrome |
| SMP | Safety Monitoring Plan |
| SOC | System Organ Class |
| SOCE | Store-operated calcium entry |
| $SpO_2$ | Oxyhemoglobin percent saturation |
| TEAE | Treatment-emergent adverse event |
| VTBI | Volume to be infused |
| WOCBP | Women of Child-Bearing Potential |

#### 1 INTRODUCTION

## 1.1 **COVID-19**

COVID-19 is a disease caused by a novel beta-coronavirus, designated SARS-CoV-2, which is in the same subgenus as the severe acute respiratory syndrome (SARS) virus. It was initially identified as the cause of a cluster of pneumonia cases in Wuhan, a city in the Hubei Province of China. It rapidly spread, resulting in an epidemic throughout China, followed by a worldwide pandemic. Person-to-person spread of SARS-CoV-2 is thought to occur mainly through close range contact via respiratory droplets but cases suggesting long-range airborne and fecal-oral transmission have been reported. The potential to transmit SARS-CoV-2 begins prior to the development of symptoms, is highest early in the course of the disease, and transmission after 7 to 10 days of illness is unlikely.

In a report from the Chinese Center for Disease Control and Prevention that included 44,672 confirmed infections, 81% of cases were mild and without pneumonia; 14% were severe with dyspnea, hypoxia, or >50% lung involvement on imaging within 24 to 48 hours; and 5% were critical with respiratory failure, shock, or multi-organ dysfunction The case-fatality rate was 2.3% with older age being associated with increased mortality. The case-fatality rate in critically ill patients was 49% (Wu and McGoogan 2020) but mortality may be decreasing as the pandemic progresses (Vahidy et al., 2020).

The pathophysiology of lung disease in COVID-19 has been described in two patients who underwent lung lobectomies for adenocarcinoma and were retrospectively found to have had COVID-19 at the time of the operation (Tian et al., 2020). Pathologic findings from these two patients were consistent with the exudative phase of ALI with edema and prominent proteinaceous exudates, vascular congestion, and inflammatory clusters with fibrinoid material and multinucleated giant cells. Hyaline membrane formation had not yet occurred in either of these two cases. In an autopsy series, severe endothelial injury and widespread pulmonary thrombosis with microangiopathy was noted (Ackermann et al., 2020).

Treatment for patients with mild disease is isolation in an outpatient setting with a focus on prevention of transmission to others. Severe disease warrants supportive care in the hospital with oxygen and ventilatory support as needed. Dexamethasone has been recommended as standard of care for patients with COVID-19 who are receiving supplemental oxygen only or are on mechanical ventilation. Remdesivir has received emergency use authorization in the United States for the treatment of COVID-19. Expert societies have recommended routine pharmacological venous thromboembolism prophylaxis. No specific therapies for the respiratory complications of COVID-19 exist and investigational agents are currently being studied.

For patients on invasive mechanical ventilation, low tidal volume ventilation (LTVV) is encouraged with prone ventilation the next step for patients who fail to achieve adequate oxygenation with LTVV. Additional options to consider for patients in whom prone ventilation fails to provide adequate oxygenation include high PEEP strategies and extracorporeal membrane oxygenation (ECMO).

### 1.2 Overview of CM4620

CM4620 is a potent and selective inhibitor of CRAC channels. CRAC channels are composed of the pore-forming plasma membrane protein Orai1 and the calcium-sensing ER gating-protein STIM1. Low levels of calcium within the ER cause the STIM1 protein to oligomerize and move to locations closely apposed to Orai1. When STIM1 binds to Orai1, the Orai1 Ca<sup>2+</sup> pore opens, permitting entry of extracellular calcium into the cell through the CRAC channel. This process is referred to as store-operated calcium entry (SOCE) and evidence suggests that SOCE through CRAC channels plays a critical role in the degradation and necrosis of pancreatic acinar cells in patients with acute pancreatitis.

The potential for CM4620 to inhibit CRAC channels was investigated by measuring the electrophysiological current ( $I_{CRAC}$ ) associated with calcium entry through CRAC channels in HEK293 cells stably expressing recombinant human Orai1/STIM1. Cellular recordings were performed using the whole-cell patch clamp method. Measurements of  $I_{CRAC}$  were made after the addition of extracellular 10 mM calcium chloride and subsequent administration of CM4620 at concentrations of 0.001, 0.01, 0.1, and 1  $\mu$ M. CM4620 was able to inhibit  $I_{CRAC}$  in a concentration-dependent manner, producing a mean 50% inhibition ( $I_{C50}$ ) value of 119 nM. Rapid and complete inhibition was achieved at 1  $\mu$ M of CM4620. Evaluations were performed to further elucidate the site of action of CM4620. A mutation in Orai1 (Orai1-V102C) is known to produce constitutively active CRAC channels without the need for STIM1. In this evaluation, successive concentrations of CM4620 produced nearly complete inhibition of the STIM1-independent  $I_{CRAC}$ , indicating that Orai1 is a major site of action of the compound.

# 1.3 Pre-Clinical Development of CM4620

## 1.3.1 Pre-Clinical Safety and Toxicology Studies

Safety pharmacology studies conducted in rats indicated no CM4620-induced adverse effects on central nervous or respiratory systems. Dose-limiting adverse clinical and cardiovascular effects were noted in a single telemetered cynomolgus monkey dosed at 25 mg/kg IV with Auxora. Cardiovascular data at lower doses (1, 3 and 10 mg/kg) showed transient, non-dose-related, slight-to-moderate increases in systolic/diastolic arterial blood pressures and negative chronotropic effects (mild and non-adverse) at all doses and in placebo treated animals.

Repeat-dose toxicity studies conducted in both rats and monkeys showed no observable adverse effect levels (NOAELs) of 25 mg/kg/day and 3 mg/kg/day, respectively. In vitro genetic toxicity studies were negative in the Ames bacterial reverse mutation assay and weakly positive/equivocal in a micronucleus assay conducted in human peripheral blood lymphocytes. A subsequent in vivo micronucleus study conducted in rats involving two different endpoints (bone marrow micronucleus and liver Comet assays) showed no evidence of DNA reactivity. Based on the results of the complete battery of genotoxicity testing, the weight of evidence indicates that CM4620 is neither mutagenic nor clastogenic. Hemolysis testing concluded that CM4620 placebo was compatible with human plasma and non-hemolytic in human blood. Specific local tolerance studies to examine irritation/inflammation at the injection site were not performed, but no evidence of compound-related or vehicle-related local irritation was observed in the repeat-dose toxicity studies in rat and monkey. Finally, in vitro 3T3 results indicated that CM4620 is potentially phototoxic, so appropriate precautions are being taken in clinical trials.

## 1.3.2 Preclinical Efficacy Studies

Support for the idea that CRAC channel inhibition could be useful in the treatment of lung injury comes from preclinical data examining the effects of BTP2, a widely used research CRAC channel inhibitor, as well as Auxora. BTP2 was shown to attenuate lipopolysaccharide-induced lung injury in mice and ventilator-induced lung injury in rats. Using a rat model of acute pancreatitis (AP), intravenous (IV) infusion of Auxora was noted to decrease lung myeloperoxidase activity (i.e., neutrophil infiltration) and mRNA levels of the pro-inflammatory cytokines TNF $\alpha$  and IL-6. Finally, knockdown of Orai1 in mice, which reduces CRAC channel activity, inhibited TNF $\alpha$ -induced cytokine expression (including IL-6) and myeloperoxidase activity in lung tissue.

Potential efficacy of CM4620 in treating acute lung injury was established in three diverse in vivo models of AP that cause both pancreatic damage and lung inflammation (TLCS-induced, FAEE-induced, and caerulein-induced acute pancreatitis models). Myeloperoxidase activity within lung tissue, as well as trypsin activity, myeloperoxidase activity and histopathological indices (edema, inflammatory cell infiltration, vacuolization, and necrosis) in pancreas tissue, were all markedly reduced following a single IP dose of CM4620 in the mouse caerulein-induced pancreatitis model, two IP doses of CM4620 in the mouse TLCS-induced and FAEE-induced pancreatitis models, and one 4-hour IV infusion of CM4620 Nanoemulsion (the intended clinical dosage form, route of administration and infusion duration) in the rat caerulein-induced pancreatitis model. The timing of CM4620 administration relative to induction of pancreatitis was investigated in the TLCS-induced and FAEE-induced pancreatitis models, and the results suggested that CM4620 may be more effective in minimizing pancreatic injury and subsequent downstream events if it is administered early in the course of disease, although later administration retains effectiveness in halting disease progression. The timing of administration for prevention or treatment of lung injury was not investigated.

# 1.4 Clinical Development of Auxora

# 1.4.1 Single Ascending Dose and Multiple Ascending Dose Studies

CalciMedica has conducted two Phase 1 studies of Auxora in healthy subjects: a single ascending dose (SAD) study (CM4620-101) and a multiple ascending dose (MAD) study (CM4620-102). In CM4620-101 (Table 1), 32 healthy subjects were enrolled in five groups and randomized in a 3:1 ratio to receive a single dose of active versus placebo. The dose levels for each group are noted in Table 1. The dose volume of the emulsion was fixed at 1.3 mL/kg for all subjects in the SAD study groups, and Auxora or placebo was administered via a 4-hour IV infusion.

**Table 1. SAD (CM4620-101)** 

| Group | Active Treatment | Number of Active<br>Treatment Subjects | Number of Placebo<br>Treatment Subjects | IV Dose Volume<br>(mL/kg) |
|---|---|---|---|---|
| 1 | 0.1 mg/kg | 6 | 2 | 1.3 |
| 2 | 0.24 mg/kg | 3 | 1 | 1.3 |
| 3 | 0.48 mg/kg | 3 | 1 | 1.3 |
| 4 | 1.0 mg/kg | 6 | 2 | 1.3 |
| 5 | 2.1 mg/kg | 6 | 2 | 1.3 |

Of the 32 enrolled subjects, there were no serious adverse events (SAE) or adverse events (AE) classified as moderate or severe in intensity. There were three clinical AEs that were all classified as mild in intensity. Two of the AEs were considered possibly related and one was considered unlikely or unrelated to study treatment. In each case, no action was taken with respect to study treatment because of the AEs. No laboratory abnormalities were observed that were considered clinically significant. There were vehicle-related increases in serum triglyceride and cholesterol levels noted in some subjects that returned to baseline within 24 hours. There was no evidence of any sustained treatment related increase in systolic or diastolic blood pressure. In addition, cardiac function, monitored by continuous electrocardiographic recording and serial biomarker testing, showed no evidence of any treatment related effect on heart rate, QTcF, cardiac troponin-T or B-type natriuretic peptide levels.

In the SAD study (CM4620-101), interim non-compartmental pharmacokinetic (PK) analysis indicates that CM4620 likely distributes to three compartments. Plasma concentrations of compound rise steadily during the 4-hour infusion, with T<sub>max</sub> achieved at the end of infusion (4 hours). After the end of infusion, there is a rapid and prominent distribution phase followed by a prolonged period of residual drug levels. The terminal elimination phase has not yet been fully characterized as it appears to be much longer than was anticipated based on pre-clinical PK data in mouse, rat, dog and monkey. Plasma concentrations during the terminal phase are approximately 5% of C<sub>max</sub> values and, as indicated above, to date there have been no clinically significant AEs reported during this phase. Plasma exposures, defined by AUC<sub>0-24h</sub>, appear to be dose-proportional and reached a maximum of 6710 ng\*h/mL in Group 5, which is 4.3-fold below the mean AUC<sub>24h</sub> in monkey at the NOAEL (29,000 ng\*hr/mL).

In the MAD study (Table 2) of Auxora (CM4620-102), subjects in the first group were randomized to receive a single dose of active treatment, 0.50 mg/kg, versus placebo for seven consecutive days. Eight healthy subjects were enrolled in the first group, with five receiving active treatment and three receiving placebo. One of the subjects received placebo at the maximum dose volume of emulsion, 1.3 mL/kg, for 7 days, whereas all others were dosed on a weight-based adjustment of dose volume. There were no SAEs and no AEs classified as moderate or severe in intensity. There were 15 clinical AEs that were all classified as mild. In each case, no action was taken with respect to study treatment because of the AEs. No laboratory abnormalities were observed that were considered clinically significant.

**Table 2.** MAD (CM4620-102)

| Group | Active Treatment<br>Daily for 7 days | | | IV Dose Volume<br>(mL/kg) |
|---|---|---|---|---|
| 1 | 0.5 mg/kg | 5 | 3 | 0.3125a |
| 2 | 1.0 mg/kg | 6 | 2 | 0.625 |

a one placebo patient received maximum dose volume of 1.3 mL/kg

Subjects in the second group of CM4620-102 were randomized to receive a single dose of active treatment, 1.0 mg/kg, versus placebo for seven consecutive days. Eight healthy subjects were enrolled in the second group, with six receiving active treatment and two receiving placebo for seven consecutive days. There were no SAEs and no AEs classified as moderate or severe in

intensity. There were three AEs that were all classified as mild in intensity. In each case, no action was taken with respect to study treatment because of the AEs. No laboratory abnormalities were observed that were considered clinically significant.

There were vehicle-related increases in serum triglyceride noted in some subjects in both groups with levels returning to baseline within 24 hours. Cholesterol levels accumulated in some subjects in both groups with daily dosing, but the increases were not considered clinically significant and were related to the vehicle. Thus, the largest rise in cholesterol levels was in the subject who received placebo at the maximum dose volume of emulsion. The rise in cholesterol is believed to be due to the release of tissue cholesterol induced by the lecithin in the emulsion (Byers et al., 1962), was noted in the pre-clinical studies in monkeys, and was reversible with cessation of dosing. There was no evidence of any sustained treatment related increase in systolic or diastolic blood pressure. In addition, cardiac function, monitored by continuous electrocardiographic recording and serial biomarker testing, showed no evidence of any sustained treatment related effect on heart rate, QTcF or B-type natriuretic peptide levels.

Non-compartmental PK analysis of Group 1 in CM4620-102 (0.5 mg/kg) indicates that CM4620 accumulated in plasma, with a 2.6-fold increase in systemic exposure (AUC<sub>24h</sub>) on Day 7 compared to Day 1 of dosing, consistent with modeling simulations. C<sub>max</sub> accumulated 1.6-fold (geometric mean of 363 ng/mL on Day 7). The geometric mean of the AUC<sub>24h</sub> on Day 7 was 3190 ng\*hr/mL, which is 9.1-fold below the NOAEL AUC<sub>24h</sub> in monkey (29,000 ng\*hr/mL). PK analysis of Group 2 in CM4620-102 (1.0 mg/kg) indicates that CM4620 accumulated in plasma, with a 2.6-fold increase in AUC<sub>24h</sub> on Day 7 compared to Day 1 of dosing, consistent with modeling simulations. C<sub>max</sub> accumulated 1.4-fold (geometric mean 637 ng/mL on Day 7). The geometric mean of the AUC<sub>24h</sub> on Day 7 was 6830 ng\*hr/mL, which is 4.2-fold below the NOAEL AUC<sub>24h</sub> in monkey (29,000 ng\*hr/mL). After the end of 7 days of infusion, there remained a prolonged period of residual drug levels in both MAD groups that remained significantly lower than the C<sub>max</sub> on Day 7. A 3<sup>rd</sup> group of healthy subjects in the MAD was not dosed, despite the benign safety profile, because of the prolonged period of residual drug levels noted in the previous groups of healthy subjects.

Subjects in Groups 4 and 5 of the SAD study and Groups 1 and 2 of the MAD study who received CM4620 were followed for 1 year in a long-term extension study to assess for adverse events and serious adverse events. In addition, PK levels were drawn in all 4 groups on Day 270 to further characterize the terminal phase and the prolonged period of residual drug level. There were no serious adverse events and no adverse events rated moderate or severe in intensity in subjects followed for 365 days.

A population PK model was built using the data from the SAD and MAD studies. The model suggested three compartments for distribution as well as gender and body weight-dependent differences in exposures. The model showed that females have a higher volume of distribution compared to males, potentially explaining the lower plasma AUC<sub>24h</sub> values versus males, and that patients with higher body weights will have a lower AUC. The model was then used to identify the dosing regimens for the first and second phases of the open-label study described below.

# 1.4.2 Open Label Study in Patients with Acute Pancreatitis with Accompanying SIRS and Hypoxemia (CM4620-201)

CalciMedica has conducted a Phase 2, open-label, dose-response, multi-center study of Auxora in patients with AP and accompanying SIRS and hypoxemia (CM4620-201). One patient was randomized having SIRS alone at Screening. The primary objective of the study was to evaluate safety and tolerability; the secondary objective was to evaluate efficacy and the PK profile of Auxora.

The study consisted of 2 phases; the Initial Phase consisted of 2 concurrently enrolled cohorts and the Second Phase consisted of 2 concurrently enrolled cohorts. In total, it was planned to have 4 Cohorts containing 24 adult male and female patients with AP and accompanying SIRS and hypoxemia. In the Initial Phase, 4 female patients were to be randomized in a 3:1 ratio to receive Auxora + Supportive Care (SC) or SC alone (Cohort 1). Concurrently, 4 male patients were to be randomized in a 3:1 ratio to receive Auxora + SC or SC alone (Cohort 2). Doses were to be 1.0 mg/kg on Day1 and 1.4 mg/kg daily on Days 2, 3 and 4 (low dose regimen). In the Second Phase, 8 female patients were to be randomized in a 3:1 ratio to receive Auxora + SC or SC alone (Cohort 3). Concurrently, 8 male patients were to be randomized in a 3:1 ratio to receive Auxora + SC or SC alone (Cohort 4). Planned doses for both Cohorts 3 and 4 were to be 2.08 mg/kg daily on Days 1 and 2 and 1.6 mg/kg daily on Days 3 and 4 (high dose regimen).

The decision to start Cohort 3 in the Second Phase was made after CalciMedica reviewed the available efficacy, safety and tolerability data from Cohort 1 and discussed this with the Principal Investigator (PI). In addition, the data was sent to the FDA for review. At this point, a decision was made to administer patients in Cohort 3 with the same dose level and schedule as in Cohort 1, as efficacy was observed in Cohort 1. Cohort 3, therefore, received the same dose level and schedule as Cohort 1, 1.0 mg.kg on Day1 and 1.4 mg/kg daily on Days 2, 3 and 4. The decision to start Cohort 4 in the Second Phase of the study was made after CalciMedica reviewed the available efficacy, safety and tolerability data from Cohort 2 and discussed this with the Principal Investigator. The data from Cohort 2 was also sent to the FDA for review. Cohort 4, therefore, received the original planned dose level and schedule; 2.08 mg/kg daily on Days 1 and 2 and 1.6 mg/kg daily on Days 3 and 4.

The first infusion of Auxora was started within 6 (up to 8) hours of the patient or LAR providing informed consent and was administered as a continuous IV infusion over 4 hours. Subsequent infusions were to be started every 24 hours (± 1 hour) from the start of the first infusion. In patients receiving Auxora+SC (all doses), there were 9 patients of 14 patients (64%) who did not receive all 4 scheduled doses, 7 of 9 patients because of rapid clinical improvement leading to early discharge and 2 of 9 patients because of study drug discontinuation. Five of 8 patients (63%) receiving the low dose regimen+SC and 4 of 6 patients (67%) receiving the high dose regimen+SC did not receive all 4 doses of Auxora.

The demographic information and baseline characteristics for the patients enrolled in the study are noted in Table 3.

Table 3. Demographics and Baseline Characteristics of Patients in CM4620-201

| Treatment | Auxora+SC<br>low dose regimen<br>(N = 8) | Auxora+SC<br>high dose regimen<br>(N = 6) | Auxora+SC<br>TOTAL<br>(N = 14) | SC Alone (N = 7) |
|---|---|---|---|---|
| Median Age (years) | 55 | 43.5 | 50.5 | 54 |
| Min, Max | 26, 66 | 37, 55 | 26, 66 | 40, 72 |
| Gender, n% | Female 5 (63%) | Female 0 | Female 5 (36%) | Female 4 (57%) |
| | Male 3 (38%) | Male 6 (100%) | Male 9 (64% | Male 3 (43%) |
| Race, n% | Asian 1 (13%) | Asian 0 | Asian 1 (7%) | Asian 0 |
| | Black 1 (13%) | Black 2 (33%) | Black 3 (21%) | Black 3 (43%) |
| | White 6 (75%) | White 4 (67%) | White 10 (71%) | White 4 (57%) |
| Median Weight (kg) | 86 | 92.8 | 87.5 | 93.1 |
| Min, Max | 56.2, 108.9 | 84.8, 113.8 | 56.2, 113.8 | 59, 108.9 |
| BMI (kg/m²) | 31.6 | 28.9 | 30.3 | 34 |
| Min, Max | 22, 44.4 | 25, 38.2 | 22, 44.4 | 23.8, 41.6 |
| Hx Type 2<br>Diabetes Mellitus | 2 (25%) | 1 (17%) | 3 (21%) | 1 (14%) |
| Hx Hypertension | 4 (50%) | 4 (67%) | 8 (57%) | 6 (86%) |

The primary objective of this study was to assess the safety and tolerability of Auxora in patients with AP and accompanying SIRS and Hypoxemia. In this study, the low dose regimen+SC and the high dose regimen+SC were well tolerated in patients with AP and SIRS, with no evidence of untoward safety or tolerability findings.

Treatment-emergent AEs (TEAEs) were reported in 7 of 8 patients (88%) receiving the low dose regimen+SC, 5 of 6 patients (83%) receiving the high dose regimen+SC, and 3 of 7 patients (43%) receiving SC alone. Severe TEAEs were reported in 0 of 8 (0%) patients receiving the low dose regimen+SC, 2 of 6 (33%) receiving the high dose regimen+SC, and 2 of 7 (29%) receiving SC alone. There were 3 TEAEs in 2 patients leading to discontinuation of the study drug. Both patients received the high dose regimen+SC.

Two different TEAE preferred terms were reported in 2 or more patients receiving the low dose regimen+SC: Hypokalemia in 2 of 8 patients (25%) and Headache in 2 of 8 patients (25%). Three different TEAE preferred terms were reported in 2 or more patients receiving the high dose regimen+SC: Malnutrition, Confusional State and Acute Respiratory Distress Syndrome were each reported in 2 of 6 patients (33%). There were no TEAE preferred terms reported in 2 or more patients receiving SC alone.

There was 1 TEAE of Chromaturia in a patient receiving the high dose regimen+SC for which the causality was considered Possible. There were no other TEAEs, for which the causality was considered Possible, Probable or Definite.

SAEs were reported in 2 of 8 patients (25%) receiving the low dose regimen+SC, 1 of 6 patients (17%) receiving the high dose regimen+SC and 2 of 7 patients (29%) receiving SC alone. There was 1 death during the study. This patient, who received the high dose regimen+SC, experienced an SAE of Hypoxic-Ischemic Encephalopathy for which the outcome was fatal. The SAE was

considered severe and the outcome was designated recovered/resolved with sequelae. Causality was considered to be Unrelated.

There were no untoward changes in vital signs, oxygenation, and laboratory values associated with treatment with either the low dose or high dose regimen of Auxora.

# 1.5 Pharmacodynamic and Pharmacokinetic Study in Patients with Acute Pancreatitis (CM4620-202)

In Study CM4620-202, A Pharmacodynamic and Pharmacokinetic Study of Auxora in Patients with Acute Pancreatitis, patients with AP (regardless of the presence of SIRS and/or hypoxemia) were administered a single IV infusion of 2.08 mg/kg Auxora and blood, plasma and serum were collected for analysis. It was planned to initially enroll 5 patients and then to enroll an additional 4 patients as needed. Ultimately, 7 patients were screened for the study, and all 7 enrolled in and completed the study. On Days 1 and 2, blood and plasma samples for PD and PK analyses, respectively, were obtained 30 minutes after completing the administration of Auxora and 24 hours from the start of the administration of Auxora. In patients hospitalized at Day 5 and 10, blood and plasma samples were obtained; if discharged earlier, samples were obtained at the time of discharge. After discharge, patients returned to the hospital on Day 30 to provide final blood and plasma samples.

Of the 7 patients, 5 (71%) were male and 2 (29%) were female. The median (min, max) age in all 7 patients was 42 (29, 54) years. The age range was 38 to 54 years in males and 29 to 35 years in females. The weight range was 49.4 to 102.1 kg and the BMI range was 19.3 to 32.2. Of the 7 patients, 4 (57%) were black or African and 3 (43%) were white. There were no (0%) Hispanic or Latino patients enrolled in the study. The cause of AP was alcohol in 5 of the 7 patients, hypertriglyceridemia in 1 of the 7, and unknown in the other.

A total of 3 patients experienced 7 TEAEs during the study. One (1) patient experienced a TEAE of Melena and a TEAE of bursitis, 1 patient had a TEAE of Pancreatitis Acute (which was also an SAE), and 1 patient experienced TEAEs of Pneumonia, Alcohol Withdrawal Syndrome, Pyrexia and Respiratory Distress (which was also an SAE). Of the 7 TEAEs, there were 3 mild, 2 moderate and 2 severe TEAEs. The 2 severe TEAEs (Pancreatitis Acute and Respiratory Distress) were also SAEs. The causality of the 7 TEAEs to Auxora was Unrelated for 5 TEAEs and Unlikely for 2 TEAEs.

# 1.6 Study in Severe Covid-19 Pneumonia (CM4620-204)

A double-blind, randomized controlled study in patients with severe Covid-19 pneumonia, characterized by the need for low-flow or high-flow oxygenation and a P/F ratio ≤300, is currently being conducted (CM4620-204). Part 1 of the study was a randomized open-label comparison of Auxora to standard of care. 30 patients were enrolled in Part 1, 26 patients receiving low-flow oxygen and 4 patients receiving high-flow oxygen. Of the 26 patients receiving low-flow oxygen, 17 patients were randomized to Auxora and 9 to standard of care. Of the 4 patients receiving high-flow oxygen, 3 were randomized to Auxora and 1 to standard

of care. Across both arms, 15 patients (75%) receiving Auxora had ≥1 AE and six patients (30%) had ≥1 SAE. Site investigators judged three AEs, each occurring in three different patients, as being related to the administration of Auxora: an episode of itching, an increase in alkaline phosphate, and a rash. They were all considered mild by the investigators and resolved. None of the reported SAEs were determined to be related to the administration of Auxora. Among patients receiving standard of care, eight (80%) had ≥ 1 AE and five (50%) had ≥ 1 SAE. There was no difference in AEs related to infections in the Auxora group when compared to standard of care (30% in each group). Two patients (10%) treated with Auxora and two patients (20%) receiving standard of care died while hospitalized between 10 and 17 days after randomization. Patients receiving low flow oxygen and treated with Auxora were noted to have a shorter median time to recovery, decreased need for invasive mechanical ventilation, and greater clinical improvement than patients receiving standard of care. A composite outcome of death or mechanical ventilation occurred less frequently in patients treated with Auxora.

Given the favorable safety profile and signals of efficacy, enrollment in the open-label study was halted, and the study was transitioned to Part 2 a double-blind RCT with matching placebo. The study is currently being conducted across multiple sites in the United States.

## 1.7 Rationale for Current Study and Selected Doses

The rationale for this study is to determine the optimal dose for use in patients with critical COVID-19 pneumonia based on pharmacodynamic markers obtained by BAL. Previous studies have randomized patients with severe COVID-19 pneumonia and acute pancreatitis with accompanying SIRS and hypoxemia who were not on a mechanical ventilator at the time of the initial infusion of Auxora. It remains necessary to determine if Auxora is an effective therapy in patients with a greater degree of diffuse alveolar damage and already requiring mechanical ventilation at the time of the initial infusion of Auxora. The selected dose may then be studied in patients with ARDS due to a variety of causes including bacterial pneumonia.

In the initial study of CM4620 in patients, CM4620-201, the low dose regimen provided the same Cmax as the highest dose in the SAD and the total exposure in the MAD was compressed into 4 days instead of 7 days of dosing. In Cohort 4, male patients received a higher dose regimen that resulted in a 30% increase in total exposure without an increase in SAEs. PK modeling from plasma levels in CM4620-201 and CM4620-202, along with analysis of the time course of IL-6 decrease, lead to the decision to study 3 doses in CM4620-204. In Part 1, it appears that patients with initial P/F ratios less than 100 treated with Auxora may have benefited from additional dosing. Therefore, this study will be undertaken to assess the changes in pharmacodynamic measures of T cell activation using initially the dose regimen from CM4620-204, then the high dose regimen from CM4620-201, and then finally, a dose regimen with 5 days of Auxora infusion.

Results of the PD *ex vivo* blood assay of lymphocyte function in Study CM4620-202 indicated that when 2.08 mg/kg of Auxora was administered, at or near the C<sub>max</sub>, CRAC channel-dependent stimulated IL-2 secretion was inhibited by approximately 57%. The inhibitory effect of Auxora dissipated over the next 1-2 days, demonstrating pharmacological reversal. This result suggests that long-term immunosuppression is unlikely to result from therapy with Auxora. Patients will be followed for 30 days to ensure that long term adverse events are collected.

#### 2 OBJECTIVES AND ENDPOINTS

## 2.1 Primary Objective

 To assess the pharmacodynamic response of bronchoalveolar lavage (BAL) T cell/monocyte subsets and chemokine release to various doses of Auxora in patients with critical COVID-19 pneumonia

## 2.2 Secondary Objectives

- To assess the safety and tolerability of Auxora in patients with critical COVID-19 pneumonia
- To determine the serum and BAL pharmacokinetic profile of Auxora in patients with critical COVID-19 pneumonia

## 2.3 Endpoints

- Pharmacodynamic endpoint:
  - Proportion of immune cells in BAL fluid (specifically: Tregs, CD4 and CD8 T cells, B cells, NK cells, alveolar macrophages monocytes, and neutrophils). T cell activation will also be assessed via flow cytometry by assessing surface expression of HLA-DR and CD127.
  - Activation of all immune cell types will be assessed using integrative analysis of single cell RNA sequencing on all subjects across all time points. After demultiplexing reads will be aligned to a hybrid genome containing human (GRCh38) and SARS-CoV-2 (NC\_045512.2) reference genomes. Resulting cell-by-gene matrices from all samples will be normalized using sctransform algorithm and integrated using BBKNN or scVI/scANVI approach followed by Leiden clustering, identification of marker genes for each cluster and assigning cell type identity to clusters (for details see Grant et al., 2021). It will be assessed whether treatment with Auxora resulted in emergence of the new clusters/cell types/cell states and markers characterizing these newly emergent populations will be evaluated. For homologous cell types differential genes expression analysis will be performed between Auxora- and placebo-treated subjects, split by time-points. The impact of Auxora treatment on detection of SARS-CoV-2 positive and negative strand RNA in infected cells will also be assessed. Differential gene expression will be performed on per-cluster level and using multilevel statistics (percluster and per subject level, to assess biological variability within the group).

## • Efficacy endpoint

- o All-Cause Mortality at Day 60
- o Number of Days on Mechanical Ventilation after randomization
- o Number of Days in the Hospital after randomization
- o Number of Days in the ICU after randomization

## • Safety endpoints

- o Pre-defined changes in cardiac conduction
- The incidence of TEAEs and SAEs
- o The intensity and relationship of TEAEs and SAEs
- o Mortality at Day 30

#### 3 INVESTIGATIONAL PLAN

## 3.1 Study Design

This will be a single-blind study where the patient will not know if they are receiving Auxora or Placebo. The first 4 patients will be enrolled in Cohort 1 and randomized 3:1 to Auxora or Placebo. If dose escalation occurs, the next 4 patients will be enrolled in Cohort 2 and randomized 3:1 to Auxora or Placebo. If dose escalation continues, the next 8 patients will be enrolled in Cohort 3 and randomized 3:1 to Auxora or Placebo. The decision to escalate dosing will be made by CalciMedica in consultation with the PI after the review of safety events in Cohorts 1 and 2.

Consultation between the PI and CalciMedica will occur if any patient receiving Auxora in Cohorts 1, 2 or 3 experiences one of the cardiac conduction events listed below during the 144 hours after the Start of the First Infusion of Study Drug (SFISD):

- QTcF interval of  $\geq$  500 msec; or
- QTcF prolongation of  $\geq$  60 msec as compared to baseline; or
- Mobitz Type II second degree atrioventricular (AV) block; or
- Third degree or high grade AV block; or
- Polymorphic Ventricular Tachycardia;

If one of the listed safety events occurs in a patient who is receiving Auxora in Cohort 1 but the event is not thought to be dose limiting, 4 additional patients will be enrolled in Cohort 1 and randomized 3:1 to Auxora versus Placebo for a total of 8 patients enrolled in the cohort, 6 randomized to Auxora and 2 to Placebo. The PI and CalciMedica will consult after all 8 patients are enrolled to determine if dose escalation to Cohort 2 will occur. If one of the listed safety events occurs in a patient who is receiving Auxora in Cohort 1 and the event is dose limiting, further dosing will not occur using the planned dose regimens but may occur using a regimen that provides lower total exposure of drug.

If one of the listed safety events occurs in a patient who is receiving Auxora in Cohort 2 but the event is not thought to be dose limiting, 4 additional patients will be enrolled in Cohort 2 and randomized 3:1 to Auxora versus Placebo The PI and CalciMedica will consult after all patients are enrolled to determine if dose escalation to Cohort 3 will occur. If one of the listed safety events occurs in a patient who is receiving Auxora in Cohort 2 and the event is dose limiting, further dosing will not occur in either Cohorts 2 or 3. 4 additional patients may be enrolled in Cohort 1 and randomized 3:1 to Auxora versus Placebo. The 4 additional patients in Cohort 1 will receive a dose regimen of an initial infusion followed by continuous infusion for 48 hours.

If one of the listed safety events occurs in a patient who is receiving Auxora in Cohort 3 but the event is not felt to be dose limiting, 4 additional patients will be enrolled in Cohort 3 and randomized 3:1 to Auxora versus Placebo for a total of 12 patients enrolled in the cohort, 9 randomized to Auxora and 3 to Placebo. If one of the listed safety events occurs in a patient

who is receiving Auxora in Cohort 3 and the event is dose limiting, further dosing will not occur in Cohort 3. 4 additional patients may be enrolled in Cohort 2 and randomized 3:1 to Auxora versus Placebo. The 4 additional patients in Cohort 2 will receive a dose regimen of an initial infusion followed by continuous infusion for 72 hours.

A study physician or appropriately trained delegate will perform assessments at Screening, immediately prior to the SFISD, and then every 24 hours (±1 hours) until 240 hours after the SFISD. After 240 hours from the SFISD, the patient will be assessed q48 hours until Day 30 after the SFISD, or until discharge if earlier. Patients who are discharged before Day 25 after the SFISD will be followed-up at Day 30 (±5 days) Patients will be followed up at Day 60 (±5 days) for a safety and mortality assessment. This assessment will be conducted by phone for patients discharged prior to Day 55. The Day 60 assessment will be completed as a final inpatient safety assessment for patients who remain hospitalized or are discharged from the hospital on Days 55-59.

Fluid from a bronchoalveolar lavage (BAL) should be obtained prior to the SFISD (-12 hours) and then again 24 ( $\pm 12$ ) hours after the last infusion of study drug in Cohorts 1 and 2. In Cohort 3, BAL fluid will be obtained during the final 24 hours of the continuous infusion. BAL fluid will be used for flow cytometry, single cell RNA sequencing, and chemokine/biomarker panel. On the BAL fluid obtained from the second BAL, CM4620 levels will be determined in patients receiving Auxora.

ECGs will be performed and the QTcF will recorded daily at each assessment until 144 (+2) hours from the SFISD. If at any time QT prolongation is suspected on a cardiac monitor, a ECG will be performed and a QTcF shall be recorded. Blood specimen for PK analysis should be obtained in patients receiving Auxora.

# 3.2 End of Study

The End of Study is considered the date on which the last patient randomized completes the visit on Day 60, unless CalciMedica terminates the study early.

# 3.3 Sponsor Termination of the Study

CalciMedica intends to complete the study as outlined. CalciMedica reserves the right, however, to terminate the study at any time or for any reason including:

- A directive from the FDA
- A lack of enrollment
- A recommendation from the IDMC

#### 4 SELECTION OF PATIENTS

#### 4.1 Inclusion Criteria

All of the following must be met for a patient to be randomized into the study:

- 1. Has laboratory-confirmed SARS-CoV-2 infection as determined by polymerase chain reaction (PCR) or other commercial or public health assay in any specimen;
- 2. Moderate ARDS characterized by the following criteria:
  - o Invasive mechanical ventilation with a minimum PEEP of 5 cm H<sub>2</sub>O;
  - PaO₂/FiO₂ ≤200 that may be estimated pulse oximetry or determined by arterial blood gas;
  - No evidence of volume overload or heart failure as the sole cause of pulmonary edema;
- 3. The patient is  $\geq 18$  years of age;
- 4. QTcF interval ≤440 milliseconds;
- 5. A female patient of childbearing potential must not attempt to become pregnant for 39 months, and if sexually active with a male partner, is willing to practice acceptable methods of birth control for 39 months after the last dose of study drug;
- 6. A male patient who is sexually active with a female partner of childbearing potential is willing to practice acceptable methods of birth control for 39 months after the last dose of study drug. A male patient must not donate sperm for 39 months;
- 7. The patient is willing and able to, or has a legal authorized representative (LAR) who is willing and able to, provide informed consent to participate, and to cooperate with all aspects of the protocol.

#### 4.2 Exclusion Criteria

Patients with any of the following conditions or characteristics must be excluded from randomizing:

- 1. Expected survival or time to withdrawal of life-sustaining treatments expected to be <7 days;
- 2. ECMO:
- 3. Invasive mechanical ventilation for more than 7 days
- 4. Suspected septic shock;
- 5. The patient has a history of:
  - a. Organ or hematologic transplant;
  - b. HIV;
  - c. Active hepatitis B, or hepatitis C infection;

- 6. Current treatment with:
  - a. Chemotherapy;
  - b. Immunosuppressive medications or immunotherapy (see Section 5.3 for list of prohibited immunosuppressive medications and immunotherapy) at the time of consent;
  - c. Hemodialysis or Peritoneal Dialysis;
- 7. The patient is known to be pregnant or is nursing;
- 8. Currently participating in another study of an investigational drug or therapeutic medical device at the time of consent;
- 9. Allergy to eggs or any of the excipients in Auxora.

# 4.3 Re-Screening

A patient who fails the initial screening may be rescreened twice again within 24 hours of the original screening.

#### 5 TREATMENT OF PATIENTS

## 5.1 Overview

All patients enrolled in the study should receive care consistent with local standard of care including for ventilator management. Patients should receive conservative intravenous fluid strategies such as FACTT LITE. All patients should receive pharmacological prophylaxis to prevent the development of venous thromboembolic disease. The type and dose of prophylaxis should be determined by local standard of care.

Patients enrolled in the study should receive dexamethasone as standard of care. If patients are not receiving dexamethasone at the time of randomization, starting dexamethasone during the hospitalization should be considered. If the patient is already receiving dexamethasone at the time of randomization, dexamethasone should be continued on its established dosing schedule. The COVID-19 Treatment Guidelines Panel of the National Institutes of Health recommends using dexamethasone (at a dose of 6 mg per day, given orally or intravenously, for up to 10 days) in patients with COVID-19 who require supplemental oxygen. Before initiating dexamethasone, the potential risks and benefits of administering corticosteroids should be assessed including risks for hyperglycemia and secondary infections. At this time, it is not known whether other corticosteroids, such as prednisone, methylprednisolone, or hydrocortisone, will have a similar benefit to dexamethasone. Of note, the dose equivalencies for dexamethasone 6 mg daily are prednisone 40 mg, methylprednisolone 32 mg, and hydrocortisone 160 mg.

If patients are not receiving remdesivir at the time of randomization, starting remdesivir during the hospitalization may be considered. If the patient is already receiving remdesivir at the time of randomization, remdesivir should be continued on its established dosing schedule. The suggested dose of remdesivir for adults weighing ≥40 kg and not requiring invasive mechanical ventilation and/or ECMO is a single dose of 200 mg infused intravenously over 30 to 120 minutes on Day 1 followed by once-daily maintenance doses of 100 mg infused intravenously over 30 to 120 minutes for 4 days (days 2 through 5). If a patient does not demonstrate clinical improvement, treatment may be extended for up to 5 additional days (i.e., up to a total of 10 days). Auxora and remdesivir should not be infused at the same time but should be given sequentially.

Patients may also be considered for the administration of convalescent plasma in the study as per local standard of care.

Immunosuppressive medications or immunotherapies are prohibited in patients randomized into the study (see Section 5.3 for the list of prohibited medications). The use of dextromethorphan in patients is discouraged when enrolled in the study.

# 5.2 Discharge Criteria

Patients should remain in the hospital until all doses of study drug have been administered.

If the patient is ready to be discharged before all doses of study drug have been administered, the PI or treating physician should contact the Medical Monitor prior to discharging the patient.

## **5.3** Prohibited Medications

Any medication, with the exception of those listed below, may be given at the discretion of the PI. Medications that should not be administered during the study to patients randomized in the study include:

- Chemotherapy
- Cyclosporine, Tacrolimus
- Sirolimus, Everolimus
- Azathioprine
- Cyclosphosphamide
- Methotrexate
- Mycophenolate
- Leflunomide
- Biologics/Monoclonals: abatacept, adalimumab, alemtuzumab, anakinra, basilizimab, belimumab, bevacizumab, brodalumab, canakinumab, certolizumab, cetuximab, clazakizumab, daclizumab, eculizumab, etanercept, golimumab, infliximab, interferon, ixekizumab, muromonab, natalizumab, omalizumab, rituximab, sarilumab, secukinumab, trastuzumab, ustekinumab, vedolizumab
- Baricitinib
- Tofacitinib

# 5.4 Compliance

Only the PI or his/her appropriately trained study staff will administer study drug to patients randomized in the trial in accordance with the protocol. Study drug must not be used for any reasons other than that described in the protocol.

### 6 PROCEDURES

## **6.1** Enrollment Procedures

Up to 32 patients will be enrolled in the study sequentially into three cohorts. If a patient discontinues study drug, withdraws consent, gets extubated or dies before the second BAL is performed, they will be replaced by the enrollment of an additional patient in the cohort.

#### 6.2 Discontinuation and Withdrawal

The term discontinuation refers to a patient or PI discontinuing the administration of study drug before all doses are administered despite the patient remaining in the hospital. Patients who do not receive all doses because the treating physician discharged them from the hospital will not be considered to have discontinued study medication.

Patients have the right to discontinue the administration of study drug at any time for any reason, without prejudice to their medical care. The PI may discontinue the administration of study drug because of an adverse event or change in medical status that raises a safety concern about the patient receiving additional doses of study drug. The PI must discontinue the administration of study drug if the patient is diagnosed with a new or recurrent malignancy. If possible, the PI should contact the Medical Monitor to review the reasons for a patient's discontinuation from study drug. The PI should also record the reason for the discontinuation in the eCRF and appropriate source documents at the site. Even if the patient discontinues receiving study drug, diligence should occur to ensure that all study visits and assessments are completed.

Withdrawal refers only to the complete withdrawal of the patient from the study because of the withdrawal of consent. The PI should inform the Medical Monitor of the withdrawal of consent and record the withdrawal of consent in the eCRF and appropriate source documents at the site.

#### 7 STUDY DRUG MATERIALS AND MANAGEMENT

## 7.1 Auxora Product Description

Auxora is to be administered as an IV infusion and is supplied as a translucent, white to yellowish, sterile, non-pyrogenic emulsion containing 1.6 mg/mL of the active pharmaceutical ingredient CM4620. Auxora is supplied as a single-use glass vial. Auxora contains egg phospholipids, medium chain triglycerides, glycerin, edetate disodium salt dehydrate (EDTA), sodium hydroxide (as needed to adjust pH), and sterile water for injection (Table 4).

**Table 4. Auxora Product Information** 

| Product Name: | CM4620 Injectable Emulsion |
|---|---|
| Dosage Form: | Injectable Emulsion (Liquid) |
| <b>Concentration of CM4620</b> | 1.6 mg/mL |
| <b>Route of Administration</b> | IV |
| <b>Physical Description</b> | Translucent, non-separated, white to yellowish emulsion |
| Inactive Ingredients | Sterile Water for Injection USP, Egg Phospholipid NF (80% Phosphatidylcholine), Medium Chain Triglycerides NF, Glycerin USP, and Edetate Disodium Salt Dihydrate (EDTA) USP. Sodium Hydroxide and Hydrochloric Acid may be added to adjust the pH. |
| Manufacturer | Bioserv Corporation<br>San Diego, CA 92121 |

# 7.2 Placebo Product Description

Matching Placebo is to be administered as an IV infusion and is supplied as a translucent, white to yellowish, sterile, non-pyrogenic emulsion carrier containing no active pharmaceutical ingredient. Placebo is supplied as an 80 mL fill in a 100 mL single-use vial. Placebo contains the same ingredients as Auxora except that it does not contain CM4620.

# 7.3 Auxora and Placebo Storage

Auxora and Placebo must be maintained in a secure location with refrigerated temperature conditions of 2 to 8°C (36 to 46°F). Precaution should be taken to ensure that Auxora and the Placebo do not freeze. Temperature logs should be maintained and available during monitor review. When a temperature is noted outside the range of 2°C to 8°C lasting for 24 hours or more, or if the temperature exceeds 20°C (68°F), or is below 0°C (32°F), CalciMedica or its designee must be notified as soon as possible. The stability of Auxora and Placebo has been demonstrated to 24 months and is being evaluated for longer periods in ongoing studies.

# 7.4 Auxora and Placebo Preparation

The study pharmacist and/or designee will be responsible for the preparation and dispensation of Auxora and Placebo. Prior to administration, Auxora and Placebo both must be transferred to

a sterile container using a sterile technique. Specific details on how to prepare Auxora and Placebo, as well as the specific components that will be used to administer both Auxora and Placebo, will be provided in the Pharmacy Manual. The Pharmacy Manual will also contain tables detailing the selected dose level and volume of administration of Auxora and Placebo.

## 7.5 Auxora and Placebo Administration

In Cohorts 1, 2, and for the first infusion in Cohort 3, study drug will be administered intravenously as a continuous infusion over 4 hours (± 30 minutes). In Cohort 3, after the end of the first infusion, a 96-hour continuous infusion will commence; during the continuous infusion study drug infusion bags will be prepared daily, each diluted up to 500 mL with the addition of normal saline and each for administration continuously over 24 hours (± 30 minutes). Study drug will be administered via a bag and tubing compatible with lipid emulsions and using a 1.2-micron filter.

The Start of the First Infusion of Study Drug (SFISD) will be considered 0 hours. In Cohorts 1 and 2, study drug will again be administered at 24 ( $\pm$ 2) and 48 ( $\pm$ 2) hours from the SFISD. In Cohort 2 study drug will also be administered at 72 ( $\pm$ 2) hours from the SFISD. In Cohort 3, study drug will be administered as a continuous infusion for 96 hours after the first infusion of study drug is completed. The dose and volume of Auxora, and the volume of Placebo, that will be administered will be calculated using the patient weight obtained at the time of hospitalization or during screening. A line into a peripheral or central vein may be used for the infusion. The peripheral IV should be 20 gauge in size or larger. The peripheral IV or central line port should be dedicated when administering Auxora or Placebo other than 0.9% normal saline. Auxora and Placebo are compatible with 0.9% normal saline. The IV tubing used to administer Auxora and Placebo must contain a 1.2 micron filter. The Pharmacy Manual will contain a recommended procedure to prime the IV tubing and flush the tubing, but this may be adapted to local nursing standards. 0.9% normal saline may be used to clear the line to ensure that the volume to be infused (VTBI) is completely administered. If the administration of Auxora or Placebo is stopped because of a technical reason, such as failure of the IV site, or IV pump malfunction, the administration of Auxora or Placebo should be resumed when the technical reason is resolved, and continued at the same rate until the infusion is completed. The total amount of time for the start of infusion to end of infusion of Auxora or Placebo should be recorded.

CalciMedica may modify at any time the administered doses of Auxora or volumes of Placebo, the days of infusion, the timing of the infusion and the rate of infusion based on review of the safety and tolerability data by the IDMC. If the administration of Auxora or Placebo is stopped because of a serious adverse event that is considered to be probably or definitely related to Auxora or Placebo, the Medical Monitor must be immediately contacted.

# 7.6 Packaging and Labeling

Preparation, packaging and labeling of Auxora and Placebo will be in accordance with current Good Manufacturing Practice of Medicinal Products (GMP) guidelines. Medication labels will comply with legal requirements for labeling of investigational products in the United States.
## 7.7 Accountability, Handling and Disposal

The PI or designee will ensure that deliveries of Auxora and Placebo from CalciMedica or its designee are received by a responsible person, and such deliveries are recorded; that Auxora and Placebo are handled and stored safely and properly; that Auxora and Placebo are only dispensed to study patients in accordance with the protocol; and that unused Auxora and Placebo is returned to CalciMedica or its designee or disposed of using standard procedures approved of in advance by CalciMedica or its designee. Appropriately trained study staff will administer all doses of Auxora and Placebo. The pharmacy will maintain a record of Auxora and Placebo accountability.

#### 8 VISITS AND STUDY SPECIFIC ASSESSMENTS

### 8.1 Screening

The PI or designee must provide informed consent to the patient, or LAR, allowing the patient or LAR adequate time to consider, ask questions and receive answers, prior to agreeing to participate.

• Record the time of the patient or LAR provides informed consent

After informed consent is obtained, the following procedures are to be performed:

- Record vital signs closest to the time of assessment
- Record height and weight closest to the time of assessment
- Record results of Sars-CoV-2 testing
- Record the P/F ratio (-4 hours); it may be estimated from pulse oximetry or determined by arterial blood gas closest to the time of assessment
- Perform ECG and record QTcF interval
- Obtain serum pregnancy test in WOCBP

If the patient satisfies all of the inclusion criteria and none of the exclusion criteria, proceed to baseline assessment.

#### 8.2 Baseline Assessment

- Draw blood samples for laboratory monitoring
- Perform the BAL and obtain fluid for flow cytometry, single cell RNA sequencing, biomarker/chemokine panel, SARS-CoV-2 PCR
- Obtain blood for biomarkers/chemokines at the time of the BAL

These blood tests for laboratory monitoring may be performed on blood already drawn in the previous 12 hours prior to randomization or after randomization but prior to the start of the first infusion of study drug. After performing procedures, proceed to randomization.

#### 8.3 Randomization

• Randomize patient as per study randomization procedure.

## 8.4 Start of First Infusion of Study Drug (SFISD) 0 hour

Record concomitant medications that were administered in the 24 hours prior to the SFISD:

• For patients in Cohorts 1, 2, and 3, infuse the first dose of study drug. The SFISD should begin within 8 hours of the patient being randomized

- Record the time when the infusion of study drug starts and finishes
- At the end of infusion of Auxora, draw blood sample for PK (+30 minutes)
- For patients in Cohort 3, begin the continuous infusion of study drug that will continue for the next 96 hours and ends 100 hours after the SFISD

### 8.5 24 hours

24 ( $\pm 1$ ) hours from the SFISD:

- Record concomitant medications that were being administered in the past 24 hours
- Record vital signs closest to the time of the assessment
- Record the P/F ratio (-4 hours); it may be estimated from pulse oximetry or determined by arterial blood gas closest to the time of the assessment
- Perform ECG and record QTcF interval (-2 hours)
- Perform AE/SAE assessment
- Draw blood sample for laboratory monitoring (-12 hours)
- Draw blood sample for PK prior to the second infusion of Auxora (-2 hours) for patients in Cohort 1 and 2. For patients in Cohort 3, draw blood sample for PK 24 hours from the SFISD (±2 hours)
- For patients in Cohorts 1 and 2, start the infusion of second dose of study drug 24 hours (±1 hour) from the SFISD
  - o Record the time when the infusion of study drug starts and finishes
- For patients in Cohort 3, the continuous infusion is ongoing

### 8.6 48 hours

48 ( $\pm$ 1) hours from the SFISD:

- Record concomitant medications that were being administered in the past 24 hours
- Record vital signs closest to the time of the assessment
- Record the P/F ratio (-4 hours); it may be estimated from pulse oximetry or determined by arterial blood gas closest to the time of the assessment
- Perform ECG and record QTcF interval (-2 hours)
- Perform AE/SAE assessment
- Draw blood samples for laboratory monitoring (-12 hours)
- Draw blood sample for PK prior to third infusion of Auxora (-2 hours) for patients in Cohort 1 and 2. For patients in Cohort 3, draw blood sample for PK 48 hours from the SFISD (±2 hours)

- For patients in Cohorts 1 and 2, start the infusion of third dose of study drug 48 hours (±1 hour) from the SFISD
  - o Record the time that the infusion of study drug starts and finishes
- For patients in Cohort 3, the continuous infusion is ongoing.

#### 8.7 72 hours

72 ( $\pm$ 2) hours from the SFISD:

- Perform BAL on patients randomized to Cohort 1 ( $\pm 12$  hours)
- At time of BAL, obtain blood for biomarkers and SARS-CoV-2 PCR in patients randomized to Cohort 1 (±12 hours)
- Perform BAL on patients randomized to Cohort 3 during the final 24 hours of the continuous infusion (between 76 and 100 hours after the SFISD). At the time of BAL, obtain blood for biomarkers and SARS-CoV-2 PCR in patients randomized to Cohort 3.
- Record concomitant medications that were being administered in the past 24 hours
- Record vital signs closest to the time of the assessment
- Record the P/F ratio (-4 hours); it may be estimated from pulse oximetry or determined by arterial blood gas closest to the time of the assessment
- Perform ECG and record QTcF interval (-2 hours)
- Perform AE/SAE assessment
- Draw blood samples for laboratory monitoring (-12 hours)
- In patients randomized to Cohort 2 draw blood sample for PK (-2 hours) prior to infusion of Auxora. For patients in Cohort 3, draw blood sample for PK 72 hours from the SFISD (±2 hours)
- In patients randomized to Cohort 2, start the infusion of fourth dose of study drug 72 hours (±1 hour) from the SFISD
  - o Record the time that the infusion of study drug starts and finishes
- For patients in Cohort 3, the continuous infusion is ongoing.

#### 8.8 96 hours

96 ( $\pm$ 2) hours from the SFISD :

- Perform BAL on patients randomized to Cohort 2 (±12 hours)
- At time of BAL, obtain blood for biomarkers and SARS-CoV-2 PCR in patients randomized to Cohort 2 (±12 hours)

- Perform BAL on patients randomized to Cohort 3 during the final 24 hours of the continuous infusion (between 76 and 100 hours after the SFISD). At the time of BAL, obtain blood for biomarkers and SARS-CoV-2 PCR in patients randomized to Cohort 3.
- Record concomitant medications that were being administered in the past 24 hours
- Record vital signs closest to the time of the assessment
- Record the P/F ratio (-4 hours); it may be estimated from pulse oximetry or determined by arterial blood gas closest to the time of the assessment
- Perform ECG and record QTcF interval (-2 hours)
- Perform AE/SAE assessment
- Draw blood samples for laboratory monitoring (-12 hours)
- For patients in Cohort 3 receiving Auxora, draw blood sample for PK (+30 minutes) at the end of the continuous infusion (anticipated at 100 hours (+30 mins) after SFISD)

#### 8.9 120 hours

120 (±2 hours) from the SFISD:

- Record concomitant medications that were administered in the past 24 hours
- Record vital signs closest to the time of assessment
- Record the P/F ratio (-4 hours); it may be estimated from pulse oximetry or determined by arterial blood gas closest to the time of the assessment
- Perform ECG and record QTcF interval (-2 hours)
- Perform AE/SAE assessment
- Draw blood samples for laboratory monitoring (-12 hours)

#### 8.10 144 hours

144 (±2 hours) from the SFISD:

- Record concomitant medications that were administered in the past 24 hours
- Record vital signs closest to the time of assessment
- Record the P/F ratio (-4 hours); it may be estimated from pulse oximetry or determined by arterial blood gas closest to the time of the assessment
- Perform ECG and record QTcF interval (-2 hours)
- Perform AE/SAE assessment
- Draw blood samples for laboratory monitoring
- Draw blood sample for PK in all patients who received Auxora

## 8.11 168 hours Until Discharge or Day 30 if Earlier

Every 48 hours starting at 168 hours (±4 hours) until discharge or Day 30, whichever is earlier:

- Perform AE/SAE assessment
- If patient is extubated, record time and date of extubation
- If patient is discharged, record date of discharge, if patient was discharged to a nursing home or extended care facility, and if patient was requiring supplemental oxygen at discharge

### 8.12 Day 60 and Day 30

Patients who were discharged before Day 25 will be contacted on Day 30 ( $\pm 5$  days) for an AE/SAE assessment as well as to determine if they are receiving supplemental oxygen. For patients discharged from the hospital on Days 25-29, the final inpatient safety assessment will substitute for the Day 30 safety and mortality assessment. The Day 30 safety and mortality assessment may be conducted with an HCP.

Patients, who have been discharged from the hospital before Day 55, will be contacted on Day  $60 \ (\pm 5 \ days)$  to determine if they are receiving supplemental oxygen, experienced any symptoms suggestive of long COVID, and developed any SAEs since the Day 30 assessment. The Day 60 assessment will be completed as a final inpatient safety assessment for patients who remain hospitalized or are discharged from the hospital on Days 55-59.

## 8.13 Study Assessments

#### **8.13.1** Concomitant Medications

The name, dose and frequency of selected medications that were administered will be recorded. Generic names should be used when possible. The administration of convalescent plasma, plus the number of units administered, should be recorded as a concomitant medication.

### 8.13.2 Vital Signs

The patient's temperature, heart rate (beats per minute), systolic and diastolic blood pressures and respiratory rate (breaths per minute) closest to the time of assessment should be recorded.

#### 8.13.3 $PO_2/FiO_2$

The P/F ratio will be estimated by the table in Appendix 1 that provides an imputed value based on the SpO<sub>2</sub> and the FiO<sub>2</sub> or will be determined from a blood gas obtained as standard of care. If the patient is no longer on a ventilator, the FiO<sub>2</sub> will be estimated using Table 5.

Table 5. Conversion of O2 Flow to FiO<sub>2</sub>

| Sumplemental Overson | Estimated FiO <sub>2</sub> (%) | | |
|---|---|---|---|
| Supplemental Oxygen<br>L/min | Nasal Cannula | Face Mask | Face Mask<br>with Reservoir |
| Room Air | 21 | | |
| 1 | 24 | | |
| 2 | 28 | | |
| 3 | 32 | | |
| 4 | 36 | | |
| 5 | 40 | 40 | |
| 6 | 44 | 50 | 60 |
| 7 | | 50 | 70 |
| 8 | | 60 | 80 |
| 9 | | 60 | 90 |
| 10 | | 60 | 95 |

Adapted from Vincent et al., 2009

### 8.13.4 Laboratory Analyses

CBC with Differential, Serum Chemistries, and D-Dimer will be performed daily.

The CBC results should include absolute or percent neutrophil and lymphocyte counts. The serum chemistries should consist of results for sodium, potassium, chloride, bicarbonate, blood urea nitrogen, creatinine, glucose, calcium, phosphorus, as well as magnesium, total protein, albumin, alkaline phosphatase, alanine transaminase (ALT), aspartate transaminase (AST), total bilirubin, lactate dehydrogenase (LDH), triglycerides, and creatine kinase (CPK).

If any of the individual serum chemistries are not offered at the site it will not be performed on patients randomized in the study.

## **8.13.5 PK Samples**

Only patients who received Auxora will have blood drawn for PK samples. The date and time when the blood sample for PK analysis was drawn shall be recorded. All samples for PK analysis should be stored at -20°C (or -80°C for no more than 35 days) until shipment on dry ice to the bio-analysis laboratory.

#### **8.13.6** Blood Biomarkers and Chemokines

Cytokines and chemokines in serum and BAL fluid supernatant that will be analyzed using Milliplex Human Cytokine/Chemokine Panel II MAGNETIC Premixed 23 Plex Kit and HCP2MAG-62K-PX23 and Milliplex Human Cytokine/Chemokine MAGNETIC BEAD Premixed 41 Plex Kit, HCYTMAG-60K-PX41 (with exclusion of RANTES, PDGFA, PDGFB which require 100-times dilution of serum/BAL fluid). Both an unbiased analysis of the data using hierarchical clustering on z-score normalized cytokine/chemokine levels as well as direct

pairwise comparison of the cytokine/chemokine levels between predefined groups (Auxora vs placebo, split by specific time points) will be performed

#### **8.13.7 BAL Fluid**

SARS-CoV-2 viral RNA will be quantified in the BAL fluid collection using the Cepheid SARS-CoV-2 Influenza A/B RSV PCR assay.

In addition, BAL fluid will be processed for flow cytometry and cell sorting as described in Grant et al., 2021. Briefly, within 12 hours after collection, BAL fluid will be filtered through 70 um nylon mesh filter, cells will be pelleted by centrifugation, red blood cells will be lysed using PharmLyse buffer and white blood cell concentration and viability will be determined using AO/PI assay on K2 Cellometer instrument. Cells will be incubated with FcBlock to prevent non-specific binding followed by incubation with antibody cocktail permitting identification of Tregs, CD4 and CD8 T cells, B cells, NK cells, alveolar macrophages, monocyte and neutrophils. Stained cells will be incubated with Live/Dead dye (SYTOX Green), data will be acquired on BD FACSAria instrument. Flow cytometry data will be analyzed using FlowJo X software, specific cell types will be identified using predefined gating strategy described in Grant et al., 2021, and data will be presented as percentage from live/CD45+ cells. An unbiased analysis of the data using hierarchical clustering on z-score normalized cell type abundance as well as direct pairwise comparison of the cell type abundance between predefined groups

(Auxora vs placebo, split by specific time points) will be performed.

Live, CD45+ non-granulocytes will be sorted into 2% BSA in PBS solution, followed by wash, counting and capture for single cell RNA-sequencing using 10x Genomics 5' V2 chemistry. Followed standard single cell RNA-sequencing library preparation and quality control, libraries will be pooled in equimolar concentration and sequenced on Illumina NovaSeq 6000 (or another compatible instrument) to the depth of ~30,000 reads per cell. After demultiplexing reads will be aligned to a hybrid genome containing human (GRCh38) and SARS-CoV-2 (NC 045512.2) reference genomes. Resulting cell-by-gene matrices from all samples will be normalized using sctransform algorithm and integrated using BBKNN or scVI/scANVI approach followed by Leiden clustering, identification of marker genes for each cluster and assigning cell type identity to clusters (for details see Grant et al., 2021). It will be assessed whether treatment with Auxora resulted in emergence of the new clusters/cell types/cell states and markers characterizing these newly emergent populations will be evaluated. For homologous cell types differential genes expression analysis will be performed between Auxora- and placebo-treated subjects, split by time-points. The impact of Auxora treatment on detection of SARS-CoV-2 positive and negative strand RNA in infected cells will be assessed. Differential gene expression will be performed on per-cluster level and using multilevel statistics (per-cluster and per subject level, to assess biological variability within the group).

#### 8.13.8 Nasopharyngeal SARS-CoV-2 PCR

A nasopharyngeal swab for SARS-CoV-2 PCR will be performed contemporaneously to the BAL fluid collection. In addition, the nasopharyngeal swab for SARS-CoV-2 PCR will be performed weekly as long as viral RNA was detected in the previous sample.

#### 9 ADVERSE EVENTS

#### 9.1 Definition of Adverse Event

An adverse event (AE) is defined as any untoward medical event in a patient regardless of its causal relationship to study treatment. An AE can be any unfavorable and unintended sign (including any clinically significant medical test abnormality), symptom, or disease temporally associated with the use of study drug, whether or not it is considered related to study drug administration. Included in this definition is any newly occurring event or previous condition that has increased in severity or frequency since the administration of study drug.

A medical test abnormality (e.g., laboratory test value, vital sign recording, ECG finding, physical examination finding) will be considered clinically significant and consequently recorded as an AE only if it meets one of the following criteria:

- Induces clinical signs or symptoms
- Requires active intervention
- Requires interruption or discontinuation of study medication

#### 9.2 Definition of Serious Adverse Event

A serious adverse event (SAE) is any AE occurring at any dose and regardless of causality that:

- Results in death
- Is life-threatening
- Requires hospitalization or prolongation of existing hospitalization
- Results in persistent or significant incapacity or substantial disruption of the ability to conduct normal life function
- Is a congenital anomaly or birth defect in an offspring of a patient receiving Auxora
- Is an important medical event

The term "life-threatening" refers to an event in which the patient was at immediate risk of death at the time of the event. It does not refer to an event that hypothetically might have caused death if it were more severe.

Important medical events are those that may not need any of the criteria defined above; however, they may be considered serious when, based upon appropriate medical judgment, they may jeopardize the patient and may require medical or surgical intervention to prevent one of the other outcomes listed in the SAE definition.

Pregnancy is not considered an AE; however, information will be collected for any pregnancies that occur during study drug administration or the thirty days thereafter. Certain pregnancy outcomes will require submission as an SAE.

## 9.3 Eliciting Adverse Event Information

At every AE/SAE assessment, the patient must be asked a standard, non-directed question, such as, "how have you been feeling since your last visit?" to elicit any medically related changes in their well-being. In addition, the hospital chart and other documents relevant to patient safety must be reviewed when the patient is in the hospital.

### 9.4 Recording Adverse Events

Recording of AEs must begin after randomization. All conditions present before randomization, including untoward medical events during Screening, should be documented as medical history. Documentation shall continue until the patient dies, the patient withdraws consent, or the patient's participation in the study ends. Information to be collected includes:

- Type of event
- Date of onset
- Date of resolution
- Investigator-specified relationship to study drug and assessment of severity
- Seriousness
- Any action taken

While an AE is ongoing, changes in the severity (e.g., worsening and improving) should be noted in the source documents, but when documenting the AE, only the total duration and the greatest severity should be recorded in the case report form. AEs characterized as intermittent require documentation of onset and duration.

All AEs reported or observed during the study must be followed to resolution. Or, if not fully resolved, until the condition has stabilized, the patient dies, withdraws consent, or CalciMedica ends the trial (whichever is first).

Adverse events resulting from concurrent illnesses, reactions to concurrent medications, or progression of disease states must also be reported. Pre-existing conditions (present before the start of the AE collection period) are considered concurrent medical conditions and should NOT be recorded as AEs. However, if the patient experiences a worsening or complication of such a concurrent condition, the worsening or complication should be recorded as an AE. Investigators should ensure that the AE term recorded captures the change in condition (e.g., "worsening of...").

Each AE should be recorded to represent a single diagnosis. Accompanying signs (including abnormal laboratory test values or ECG findings) or symptoms should NOT be recorded as additional AEs. If a diagnosis is unknown, sign(s) or symptom(s) should be recorded as an AE(s).

Elective procedures (surgeries or therapies) performed to manage/treat conditions that existed prior to the patient enrolling in the trial should not be recorded as AEs but should be documented in the patient's source documents. If a planned procedure is performed early (e.g., as an emergency) because the pre-existing condition worsens, the worsening condition should be captured as an AE.

### 9.5 Assessment of Relationship to Study Drug

The Investigator must use the following classification and criteria to characterize the relationship or association of study drug in causing or contributing to the AE:

- **Unrelated**: This relationship suggests that there is no association between study drug and the reported event
- Unlikely: This relationship suggests that there is an unlikely association between study drug and the reported event
- **Possible**: This relationship suggests that treatment with study drug caused or contributed to the AE. That is, the event follows a reasonable temporal sequence from the time of study drug administration, and/or follows a known response pattern to the study drug, but could have been produced by other factors
- **Probable**: This relationship suggests that a reasonable temporal sequence of the event with study drug administration exists and, based upon the known pharmacological action of the drug, known or previously reported adverse reactions to the drug or class of drugs, or judgment based on the Investigator's clinical experience, the association of the event with study drug administration seems likely
- **Definite**: This relationship suggests a definite causal relationship exists between study drug administration and the AE, and other conditions (concurrent illness, progression/expression of disease state, or concurrent medication reaction) do not appear to explain the event

## 9.6 Assessment of Severity

The Investigator must use the following criteria to rate the intensity of the AE:

- Mild: Symptoms causing no or minimal interference with usual social and functional activities
- **Moderate**: Symptoms causing greater than minimal interference with usual social and functional activities
- Severe: Symptoms causing inability to perform usual social and functional activities

## 9.7 Reporting of Serious Adverse Events

The Investigator is responsible for reporting to CalciMedica or designee within 24 hours from the time when site personnel learn about the event, all SAEs that are observed or reported by the patient during the study (from randomization until the patient dies, the patient withdraws consent, or the patient's participation in the study ends) regardless of the relationship to study drug or clinical significance. Any additional information that becomes available later should be submitted within 1 working day of receipt. All SAEs reported or observed during the study must be followed to resolution or until the Investigator deems the event to be chronic or the patient to

be stable. CalciMedica or its designee may contact the Investigator to obtain additional information on any SAE that has not resolved at the time the patient completes the study. SAEs ongoing at database lock will be noted as such. The PIs are also responsible for informing their IRB/EC of any SAEs at their site. SAE correspondence with IRBs/ECs must be submitted to CalciMedica or its designee for filing.

A study manual will contain the details needed to report SAEs. If any questions on SAEs, contact information is as follows:

• SAE reporting email address: CalciMedicaSafety@safety-sphere.com

• SAE phone number: 844-965-1070 (toll free)

• **SAE Fax number**: 1 (833) 292-6393

CalciMedica will notify the FDA in a written safety report of any suspected adverse reaction or adverse reaction associated with the use of Auxora that is serious and unexpected.

- Suspected adverse reaction means any adverse event for which there is a reasonable possibility that the drug caused the adverse event. For the purposes of IND safety reporting, 'reasonable possibility' means CalciMedica determines that there is evidence to suggest a causal relationship between the drug and the adverse event (definite, probable, possible) regardless of the investigator's causality assessment
- Adverse reaction means any adverse event caused by a drug. Adverse reactions are a subset of all suspected adverse reactions where there is reason to conclude that the drug caused the event
- Serious, as defined in Section 9.2
- Unexpected adverse event or suspected adverse reaction refers to an event or reaction that is not listed in the investigator's brochure or is not listed at the specificity or severity that has been observed

CalciMedica or its designee will notify the FDA of any unexpected serious suspected adverse reactions associated with the use of Auxora that are fatal or life threatening as soon as possible but no later than seven calendar days after the initial receipt of the information. Initial notification will be followed by a written report within fifteen calendar days.

CalciMedica or its designee will notify the FDA of any unexpected serious suspected adverse reactions associated with the use of Auxora that are not fatal or life threatening fifteen calendar days.

CalciMedica or its designee will provide copies of any reports to regulatory agencies regarding unexpected serious suspected adverse reactions associated with the use of Auxora to the Investigators for review and submission to the IRB/EC.

The Safety Monitoring Plan (SMP) will contain specific study pause criteria for the occurrence of severe unexpected serious suspected adverse reactions associated with the use of Auxora.

In addition, the following serious adverse events that are commonly observed in this patient population will not be reported to the regulatory authority as individual expedited reports except in unusual circumstances:

- Hypoxemia and acute respiratory distress syndrome
- Oliguria and acute kidney injury
- Hypotension and shock, including septic shock
- Disseminated Intravascular Coagulation
- Venous and Arterial Thromboembolism
- Leukocytosis and Leukopenia
- Thrombocytopenia
- Lymphopenia
- Hyperbilirubinemia or Transaminitis
- Rhabdomyolysis
- Bacteremia
- Pneumonia
- Pleural Effusion
- Obtundation
- Gastroparesis and ileus

## 9.8 Suspected Pregnancy in a Woman of Childbearing Potential

A female patient of childbearing potential is a female who is not surgically sterile (no history of a bilateral salpingo-oophorectomy) and is not postmenopausal for at least 1 year.

A female patient of childbearing potential who receives study drug and is sexually active with a male partner, and a male patient who receives study drug and is sexually active with a female of childbearing potential, must be willing to use two highly effective methods of contraception (e.g., barrier methods, spermicidals, intrauterine devices, and/or hormonal contraception) for 39 months after last dose of study drug. No contraception is required if a female patient or partner has undergone a bilateral salpingo-oophorectomy.

Two of the following methods of birth control must be practiced unless a sexually active female patient or partner of childbearing potential has undergone a bilateral salpingo-oophorectomy:

- Male partner has a vasectomy for at least six months duration
- Use of an intrauterine device
- Use of hormonal contraceptives (oral, parenteral, vaginal or transdermal)

 Double barrier contraception with the male partner using a condom and the female using a contraceptive sponge, spermicidal jelly or cream or diaphragm plus spermicidal jelly or cream

The Investigator should be immediately informed if a female patient or partner of childbearing potential suspects she is pregnant up to 39 months after last dose of study drug. If the female patient is receiving study drug when discovered to be pregnant, the study drug should be immediately discontinued. If a pregnancy is confirmed, the Investigator must immediately report a pregnancy and record the event using a Pregnancy Report Form. Pregnancy is not considered an AE, but the Investigator must follow a pregnant patient or partner. The Investigator must report follow-up information regarding the course of the pregnancy, including perinatal or neonatal outcome. Infants resulting from such pregnancies should be assessed for normality at birth and should be followed for 6 months to assess for development milestones. CalciMedica or its designee may contact the Investigator to request additional information throughout the course of the pregnancy.

The following pregnancy outcomes must be considered SAEs and will require additional reporting in the eCRF and on an SAE form:

- Congenital anomaly/birth defect
- Stillbirth
- Spontaneous miscarriage

#### 10 STATISTICAL METHODS

#### 10.1 General Considerations

Sample size considerations were based on precision estimates and the ability to construct 95% confidence intervals around point estimates for pharmacodynamics endpoints with reasonable precision. Sample sizes as small as 9 patients per arm will allow for construction of 95% confidence intervals with half-widths as small as 0.77 standard deviation units.

For other assessments (flow cytometry analysis of BAL, single-cell RNA-sequencing analysis of immune cells in BAL, plasma and BAL fluid cytokines/chemokines), the study is not powered for analysis with inferential statistics.

## 10.2 Study Endpoints

Primary Pharmacodynamic endpoint:

- Proportion of immune cells in BAL fluid (specifically: Tregs, CD4 and CD8 T cells, B cells, NK cells, alveolar macrophages, monocytes and neutrophils). T cell activation will also be assessed via flow cytometry by assessing surface expression of HLA-DR and CD127.
- Activation of all immune cell types will be assessed using integrative analysis of single cell RNA sequencing on all subjects across all time points. After demultiplexing reads will be aligned to a hybrid genome containing human (GRCh38) and SARS-CoV-2 (NC\_045512.2) reference genomes. Resulting cell-by-gene matrices from all samples will be normalized using sctransform algorithm and integrated using BBKNN or scVI/scANVI approach followed by Leiden clustering, identification of marker genes for each cluster and assigning cell type identity to clusters (for details see Grant et al., 2021). It will be assessed whether treatment with Auxora resulted in emergence of the new clusters/cell types/cell states and markers characterizing these newly emergent populations will be evaluated. For homologous cell types differential genes expression analysis will be performed between Auxora- and placebo-treated subjects, split by time-points. The impact of Auxora treatment on detection of SARS-CoV-2 positive and negative strand RNA in infected cells will also be assessed. Differential gene expression will be performed on per-cluster level and using multilevel statistics (per-cluster and per subject level, to assess biological variability within the group).

Efficacy endpoints will include:

- All-Cause Mortality at Day 60
- Number of days on Mechanical Ventilation after randomization
- Number of Days in the Hospital after randomization
- Number of Days in the ICU after randomization

Safety endpoints will include:

• Pre-defined changes in cardiac conduction

- The incidence of TEAEs and SAEs
- The intensity and relationship of TEAEs and SAEs
- Mortality at Day 30

### 10.3 Analysis Sets

### 10.3.1 Pharmacodynamic and Efficacy Analysis Set

Pharmacodynamic and efficacy analyses will be based on the ITT principle. The Efficacy Analysis Set will include data from all subjects randomly assigned to study treatment. All data will be included and no subjects will be excluded because of protocol violations. For the analysis of efficacy data, subjects will be included in the treatment group according to their randomly assigned treatment.

### 10.3.2 Safety Analysis Set

The Safety Analysis Set will include data from all subjects randomly assigned to study treatment who receive any amount of Auxora or Placebo. All data will be included and no subjects will be excluded because of protocol violations.

For safety data analysis, subjects will be included in the treatment group according to the treatment they actually receive.

## 10.4 Disposition

The number and percentage (n, %) of patients screened, enrolled, treated, completed study, and discontinued (with reason) will be summarized. All screened patients will be included in the disposition analysis.

## 10.5 Analysis of Demographic and Baseline Data

Patient demographic and baseline characteristics will be summarized by mean, standard deviation, median, minimum, and maximum for continuous variables; and by counts and percentages for categorical variables.

## 10.6 PD Analysis

Primary analyses will leverage descriptive statistics to summarize the change in combined proportions of CD4, CD8, and monocytes in BAL fluid by dose arm. Point estimates and corresponding 95% confidence intervals will be reported. We will explore ANCOVA models to compare the difference in post-dose proportions by arm, adjusting for pre-dose levels. Normality assumptions will be assessed and in the event of violation of assumptions, transformations or nonparametric approaches will be considered. Subsequent pairwise comparisons of each dose

arm to placebo arm will be assessed as appropriate. Similar methods will be employed for additional flow cytometry endpoints as described above.

Exploratory analyses may also consider unsupervised methods including hierarchical clustering to further identify and visualize patterns in flow cytometry data.

Activation of all immune cell types will be assessed using integrative analysis of single cell RNA sequencing on all subjects across all time points. After demultiplexing reads will be aligned to a hybrid genome containing human (GRCh38) and SARS-CoV-2 (NC\_045512.2) reference genomes. Resulting cell-by-gene matrices from all samples will be normalized using sctransform algorithm and integrated using BBKNN or scVI/scANVI approach followed by Leiden clustering, identification of marker genes for each cluster and assigning cell type identity to clusters (for details see Grant et al., 2021). It will be assessed whether treatment with Auxora resulted in emergence of the new clusters/cell types/cell states and markers characterizing these newly emergent populations will be evaluated. For homologous cell types differential genes expression analysis will be performed between Auxora- and placebo-treated subjects, split by time-points. The impact of Auxora treatment on detection of SARS-CoV-2 positive and negative strand RNA in infected cells will also be assessed. Differential gene expression will be performed on per-cluster level (as implemented in Scanpy package) and using multilevel statistics (per-cluster and per subject level, to assess biological variability within the group, using averaged RNA expression and DESeq2 framework).

### 10.6.1 Mortality at Day 60 and Day 30

Mortality rate at Day 60 and Day 30 for each treatment group will be estimated by the Kaplan-Meier procedure.

### **10.6.2** Number of Days in the Hospital

The date of each hospital admission and discharge will be collected for each subject. The number of days when subjects are still alive and out of hospital during the first 30 Days of the study will be summarized by treatment group. We will explore nonparametric comparisons of days in hospital after randomization between arms.

### 10.6.3 Number of Days in the ICU and Days on Mechanical Ventilation

The analysis will be the same as the number of days in the hospital

## 10.7 Safety Analysis

Safety will be assessed by subject reported and Investigator observed AEs along with clinical laboratory tests (hematology and chemistries), and vital signs. Safety variables will be tabulated by treatment groups and presented for all treatment patients. Exposure to study treatments, reasons for discontinuation, deaths and causes of deaths will be tabulated. Treatment-emergent AEs (TEAEs) are defined as events that first occurred or worsened after the first dose of study

drug. TEAEs will be mapped to the appropriate System Organ Class (SOC) and Preferred Term (PT) according to the Medical Dictionary for Regulatory Activities (MedDRA).

Summaries will be provided for all AEs, AEs considered related to study treatment, SAEs, and related SAEs, AE leading to treatment discontinuation and AE leading to death as follows:

- By maximum severity
- Incidence by SOC (by severity grade and overall)
- Incidence by PT (by severity grade and overall)

Laboratory test results will be used in the summary. The lower and upper reference range values for tests from the laboratories will be used to grade the lab results to low, normal and high Shift tables will display (1) shift from baseline grade to the worst grade, and (2) shift from baseline grade to the last grade.

Vital signs will be summarized by visit using proportion of patients with each vital sign being too high or too low according to conventionally accepted vital sign normal ranges.

Concomitant medication will be coded by the WHO Drug Dictionary and summarized by Therapeutic subgroup and preferred terms, using counts and percentages. Concomitant medications are the medications taken with a start date on or after the start of the administration of study treatment, or those with a start date before the start of the administration of study treatment and a stop date on or after the start of the administration of study treatment.

Descriptive statistics will include mean, standard deviation, minimum, median, and maximum for guadecitabine and decitabine PK concentrations.

## 10.8 PK Analysis

Descriptive statistics will include mean, standard deviation, minimum, median, and maximum for PK parameters and concentrations.

The relationship between exposure and response will be assessed based on the PK data and efficacy/safety data collected in this study. The methods will include a population PK modeling approach using the sparse data collected. The details of population PK modeling and full results of the exposure response analyses will be reported in a separate document, and the summary of key findings will be included in the clinical study report.

#### 11 ADMINISTRATIVE CONSIDERATIONS

## 11.1 Monitoring of the Study

The site monitor, as a representative of CalciMedica, will closely follow the conduct of the study. The site monitor will collaborate with the study site to maintain necessary communication with the PI and his/her study staff through telephone, email, etc.. The site monitor will maintain current knowledge of each site's study activity by observing the conduct of the study at the site, reviewing study records and source documentation (remote monitoring), performing study drug accountability, reviewing the site files (i.e. regulatory documentation, training records, etc.) and discussing the conduct of the study with the PI and his/her study staff.

### 11.2 Inspection of Records

The PI, his/her study staff and the study site will provide access to all study records to assist study-related monitoring and audits, Institutional Review Board/Ethics Committee/Research Ethics Board reviews, and regulatory inspections. In the event of an audit, the PI agrees to allow CalciMedica or its representatives and relevant regulatory authorities access to all study records.

If any regulatory agency schedules an audit, the PI should promptly notify CalciMedica or its representatives and promptly forward to CalciMedica copies of any audit reports he/she receives.

## 11.3 Study Record Retention

The PI or his/her study staff must retain essential documents for at least 2 years after the last approval of a marketing application in an ICH region. They should retain these documents longer if required because of regulatory requirements or because of an agreement with CalciMedica.

## 11.4 Study Conduct: Good Clinical Practice and Declaration of Helsinki

CalciMedica will design the clinical study, shall implement it, and report it in accordance with the ICH Harmonized Guideline for Good Clinical Practice, with applicable local regulations (e.g., European Directive 2001/83/EC and US Code of Federal Regulations Title 21), and with the ethical principles laid down in the Declaration of Helsinki.

The PI agrees to conduct the study in accordance with the ICH Guideline for Good Clinical Practice, with applicable local regulations (e.g., European Directive 2001/83/EC and US Code of Federal Regulations Title 21) and with the principles of the Declaration of Helsinki. The PI must conduct all aspects of this study in accordance with all national, state and local laws or regulations.

## 11.5 Responsibilities of the Investigator and the IRB/EC

A properly constituted IRB/EC must review and approve the protocol and the proposed informed consent form before the start of the study at the site. The PI or his/her study staff must provide

CalciMedica or its designee a signed and dated statement that the IRB/EC has approved the protocol and the informed consent form before consenting patients for the study. Prior to starting the study, the PI will sign a protocol signature page confirming that he/she will conduct the study in accordance with this protocol and he/she will give CalciMedica or its designee and regulatory authorities access to all relevant data and records.

The IRB/EC chairperson or designee must sign all IRB/EC approvals and must identify the IRB/EC by name and address, the clinical protocol, and the date of approval.

The PI is responsible for obtaining reviews of the clinical research at intervals specified by the IRB/EC. The specified intervals should not exceed 1 year. The PI must supply CalciMedica or its designee written documentation of the reviews of the clinical research.

## 11.6 Confidentiality

All laboratory specimens, evaluation forms, reports, and other records will be identified in a manner designed to maintain patient confidentiality. All records will be kept in a secure storage area with limited access. Clinical information will not be released without the written permission of the patient (or the patient's legal representative) except as necessary for monitoring and auditing by CalciMedica or its designee, inspections by relevant regulatory authorities, or reviews by the IRB/EC.

The PI, all study staff and all co-workers involved in the study may not disclose or use for any purpose other than the conduct of the study any data, record or other unpublished confidential information disclosed to them for the purpose of the study. They must obtain prior written agreements from CalciMedica or its designee for the disclosure of any said confidential information to other parties.

#### 11.7 Modification of the Protocol

Any changes that arise after the approval of the protocol must be documented as protocol amendments. Amendments (substantial/non-substantial) require regulatory approval and IRB/EC approval or notification. Only after approval by CalciMedica, the PI, the IRB/EC, and if applicable the regulatory authorities, will the protocol amendments become effective. In cases when the protocol is amended to enhance patient safety, the amendment may be implemented but must be immediately submitted to the IRB/EC and regulatory authorities.

The revision number and date of the amendment will be recorded on the title page of the protocol.

The PI is responsible for informing the IRB/EC of all problems involving risks to patients. In case of urgent safety measures, CalciMedica or its designee will immediately notify the PIs and relevant regulatory authorities.

#### 11.8 Informed Consent

Because the study will be conducted under a United States Investigational New Drug Application, informed consent that is in compliance with Title 21 of the United States Code of Federal Regulations (CFR) Part 50 will be obtained from each patient or LAR before the patient enters the study or before any unusual or non-routine procedure is performed. For sites outside the United States, the signed informed consent form will be obtained in compliance with local regulations, ICH E6 (R2) and the principles of the Declaration of Helsinki.

CalciMedica or it's designee may provide to the PI or his/her study staff an informed consent form template. The informed consent form must be reviewed by CalciMedica or its designee before the PI or his/her study staff submits it to the IRB/EC. After CalciMedica or its designee review the informed consent form, the PI or his/her study staff will submit it to the IRB/EC for review and approval. If the informed consent form is revised during the course of the study, CalciMedica or its designee must agree with revisions before the PI or his/her study staff submits it to the IRB/EC. The study staff must provide CalciMedica or its designee a copy of the revised informed consent form after IRB/EC approves it. All patients or LARs affected by the revision must sign the revised informed consent form after the IRB/EC approves it.

Before enrolling in the study, each prospective patient or LAR will receive a full explanation of the study and review the approved informed consent form. Once the PI or designee is assured that the patient or LAR understands the implications of participating in the study, he/she will ask the patient or LAR to give consent for the patient to participate in the study by signing the informed consent form.

A patient may participate in the study only after providing consent using an IRB/EC approved informed consent form. A LAR of the patient may provide informed consent on behalf of the patient under conditions authorized by local laws and regulations. The patient or LAR must provide informed consent before the patient undergoes any study-specific procedures described in the protocol. The PI or designee will provide a copy of the informed consent form to the patient and/or LAR. The process of obtaining informed consent must also be documented in the patient source documents.

#### 11.9 Protocol Violations and Deviations

The PI or designee must document any protocol deviation or violation. Reporting of protocol deviations and violations to the appropriate IRB/EC is the responsibility of the PI and must follow the applicable IRB/EC guidelines.

Major protocol deviations are a subset of protocol deviations that might significantly affect the completeness, accuracy, and/or reliability of the study data or that might significantly affect a patient's rights, safety, or well-being.

If there is an immediate hazard to the patient, the PI may deviate from the protocol without prior approval from CalciMedica or its designee and the IRB/EC but must notify CalciMedica or its designee and IRB/EC of the deviation as soon as he/she is able to do so.

#### 11.10 Financial Disclosure

PIs and sub-investigators are required to document financial disclosure information prior to conducting any study procedures. In addition, the PIs and sub-investigators must provide CalciMedica or its designee with updated information if any relevant changes occur during the course of the study and for one year following the completion of the study.

Any PIs, sub-Investigators or study staff with a vested financial interest in the success of the study may not participate in the study.

### 11.11 Sponsor Obligations

CalciMedica or designee is not financially responsible for further testing/treatment of any medical condition that may be detected during Screening. In addition, CalciMedica is not financially responsible for the treatment of the patient's underlying disease.

### 11.12 Investigator Documentation

The PI will be asked to comply with ICH E6 (R2) 8.2 and title 21 CFR by providing to CalciMedica or designee the following documents:

- The IRB/EC approval of the protocol
- The IRB/EC approved informed consent form
- Any written information regarding the study that will be provided to the patient or LAR
- A Form FDA 1572, fully executed, and all updates on new fully executed Form FDA 1572 (Unless granted an exemption by the FDA and in compliance with local regulations)
- Curricula Vitae for the PI and each sub-Investigator listed on Form FDA 1572. Evidence of licensure must be noted on the Curricula Vitae or a copy of the license must be provided. The Curricula Vitae must have been updated by the PI and sub-Investigators within 3 years before study start-up to indicate that the documents are accurate and current
- Completed financial disclosure forms to allow CalciMedica or designee to submit
  complete and accurate certification or disclosure statements required under US Title
  21 CFR 54. In addition, the PI and sub-Investigators must provide to CalciMedica or
  designee a commitment to update this information promptly if any relevant changes occur
  during the course of the study and for 1 year following completion of the study
- Laboratory certifications and normal ranges for any laboratories used by the site for the conduct of the study

## 11.13 Clinical Study Insurance

CalciMedica has subscribed to an insurance policy, covering in its terms and provisions its legal liability for injuries caused to participating persons and arising out of this research that is

performed strictly in accordance with the scientific protocol as well as with applicable law and professional standards.

#### 11.14 Use of Information

All information supplied by CalciMedica to the PI and his/her study staff is privileged and confidential. The PI and his/her study staff agree to use this information to accomplish the study and not to use it for other purposes without consent from CalciMedica. Furthermore, the PI and his/her study staff are obligated to provide CalciMedica with complete data obtained during the study. The information obtained from the clinical study will be used towards the development of Auxora, and may be disclosed to regulatory authorities, other Investigators, corporate partners or consultants as required.

#### 11.15 Publications

CalciMedica Inc. reserves the right to review all planned communications and manuscripts based on the results of this study. This reservation of the right is not intended to restrict or hinder publication or any other dissemination of study results, but rather to allow CalciMedica to confirm the accuracy of the data, to protect proprietary information, and to provide comments based on information that may not yet be available to the study investigators. CalciMedica Inc. supports communication and publication of study results whatever the findings of the study. CalciMedica Inc. also encourages disclosure of any conflict of interest from all authors or investigators when manuscripts are submitted for publication.

## 11.16 Independent Data Monitoring Committee

An IDMC will be convened and will monitor safety for this study on an ongoing basis. An IDMC charter will govern the IDMC and will describe the scope of responsibilities of the IDMC. If the IDMC recommends alteration of the dosing regimen because of safety issues, the FDA and other regulatory agencies will be notified as appropriate. The IDMC responsibilities include protecting the safety of the study patients and making recommendations to CalciMedica concerning the conduct of the study.

#### 12 REFERENCES

Ackermann M, Verleden SE, Kuehnel M, Haverich A, Welte T, Laenger F, Vanstapel A, Werlein C, Stark H, Tzankov A, Li WW, Li VW, Mentzer SJ, Jonigk D. Pulmonary Vascular Endothelialitis, Thrombosis, and Angiogenesis in Covid-19. N Engl J Med. 2020;383(2):120-8. doi: 10.1056/NEJMoa2015432.

Byers SO, Friedman M, Sugiyama T. Mechanism underlying phosphatide-induced hypercholesterolemia. J Biol Chem. 1962;237:3375-80.

Fowler AA, III, Truwit JD, Hite RD, Morris PE, DeWilde C, Priday A, Fisher B, Thacker LR, 2nd, Natarajan R, Brophy DF, Sculthorpe R, Nanchal R, Syed A, Sturgill J, Martin GS, Sevransky J, Kashiouris M, Hamman S, Egan KF, Hastings A, Spencer W, Tench S, Mehkri O, Bindas J, Duggal A, Graf J, Zellner S, Yanny L, McPolin C, Hollrith T, Kramer D, Ojielo C, Damm T, Cassity E, Wieliczko A, Halquist M. Effect of Vitamin C Infusion on Organ Failure and Biomarkers of Inflammation and Vascular Injury in Patients With Sepsis and Severe Acute Respiratory Failure: The CITRIS-ALI Randomized Clinical Trial. JAMA. 2019;322(13):1261-70. doi: 10.1001/jama.2019.11825.

Grant RA, Morales-Nebreda L, Markov NS, Swaminathan S, Querrey M, Guzman ER, Abbott DA, Donnelly HK, Donayre A, Goldberg IA, Klug ZM, Borkowski N, Lu Z, Kihshen H, Politanska Y, Sichizya L, Kang M, Shilatifard A, Qi C, Lomasney JW, Argento AC, Kruser JM, Malsin ES, Pickens CO, Smith SB, Walter JM, Pawlowski AE, Schneider D, Nannapaneni P, Abdala-Valencia H, Bharat A, Gottardi CJ, Budinger GRS, Misharin AV, Singer BD, Wunderink RG, & The NU SCRIPT Study Investigators. Circuits between infected macrophages and T cells in SARS-CoV-2 pneumonia. Nature. 2021. doi: 10.1038/s41586-020-03148-w.

Tian S, Hu W, Niu L, Liu H, Xu H, Xiao S-Y. Pulmonary Pathology of Early-Phase 2019 Novel Coronavirus (COVID-19) Pneumonia in Two Patients With Lung Cancer. Journal of Thoracic Oncology. 2020. doi: 10.1016/j.jtho.2020.02.010.

Vahidy FS, Drews AL, Masud FN, Schwartz RL, Askary BB, Boom ML, Phillips RA. Characteristics and Outcomes of COVID-19 Patients During Initial Peak and Resurgence in the Houston Metropolitan Area. JAMA. 2020;324(10):998-1000. doi: 10.1001/jama.2020.15301.

Vincent JL, Rello J, Marshall J, Silva E, Anzueto A, Martin CD, Moreno R, Lipman J, Gomersall C, Sakr Y, Reinhart K, Investigators EIGo. International study of the prevalence and outcomes of infection in intensive care units. JAMA. 2009;302(21):2323-9.

Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020. doi: 10.1001/jama.2020.2648.

# Appendix 1. Imputed PaO<sub>2</sub> /FiO<sub>2</sub> Ratio

SpO<sub>2</sub>

| | SPC2 | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 0.7 | 0.75 | 0.8 | 0.81 | 0.82 | 0.83 | 0.84 | 0.85 | 0.86 | 0.87 | 0.88 | 0.89 | 0.9 | 0.91 | 0.92 | 0.93 | 0.94 | 0.95 | 0.96 |
| 0.21 | 174 | 191 | 211 | 216 | 221 | 226 | 232 | 238 | 245 | 252 | 260 | 269 | 279 | 291 | 304 | 319 | 337 | 360 | 390 |
| 0.24 | 153 | 167 | 185 | 189 | 193 | 198 | 203 | 208 | 214 | 221 | 228 | 236 | 244 | 254 | 266 | 279 | 295 | 315 | 341 |
| 0.27 | 136 | 148 | 164 | 168 | 172 | 176 | 180 | 185 | 190 | 196 | 202 | 209 | 217 | 226 | 236 | 248 | 262 | 280 | 303 |
| 0.28 | 132 | 143 | 157 | 161 | 164 | 168 | 175 | 179 | 182 | 189 | 196 | 204 | 211 | 218 | 229 | 239 | 254 | 271 | 293 |
| 0.3 | 122 | 133 | 148 | 151 | 155 | 158 | 162 | 167 | 171 | 177 | 182 | 189 | 196 | 203 | 213 | 223 | 236 | 252 | 273 |
| 0.32 | 116 | 125 | 138 | 141 | 144 | 147 | 153 | 156 | 159 | 166 | 172 | 178 | 184 | 191 | 200 | 209 | 222 | 238 | 256 |
| 0.35 | 105 | 114 | 127 | 129 | 132 | 136 | 139 | 143 | 147 | 151 | 156 | 162 | 168 | 174 | 182 | 191 | 202 | 216 | 234 |
| 0.36 | 103 | 111 | 122 | 125 | 128 | 131 | 136 | 139 | 142 | 147 | 153 | 158 | 164 | 169 | 178 | 186 | 197 | 211 | 228 |
| 0.4 | 92 | 100 | 111 | 113 | 116 | 119 | 122 | 125 | 129 | 132 | 137 | 141 | 147 | 153 | 159 | 168 | 177 | 189 | 205 |
| 0.44 | 84 | 91 | 100 | 102 | 105 | 107 | 111 | 114 | 116 | 120 | 125 | 130 | 134 | 139 | 145 | 152 | 161 | 173 | 186 |
| 0.45 | 81 | 89 | 98 | 101 | 103 | 106 | 108 | 111 | 114 | 118 | 121 | 126 | 130 | 136 | 142 | 149 | 157 | 168 | 182 |
| 0.5 | 73 | 80 | 89 | 91 | 93 | 95 | 97 | 100 | 103 | 106 | 109 | 113 | 117 | 122 | 128 | 134 | 142 | 151 | 164 |
| 0.55 | 67 | 73 | 81 | 82 | 84 | 86 | 89 | 91 | 94 | 96 | 99 | 103 | 107 | 111 | 116 | 122 | 129 | 138 | 149 |
| 0.6 | 61 | 67 | 74 | 76 | 77 | 79 | 81 | 83 | 86 | 88 | 91 | 94 | 98 | 102 | 106 | 112 | 118 | 126 | 136 |
| 0.65 | 56 | 62 | 68 | 70 | 71 | 73 | 75 | 77 | 79 | 81 | 84 | 87 | 90 | 94 | 98 | 103 | 109 | 116 | 126 |
| 0.7 | 52 | 57 | 63 | 65 | 66 | 68 | 70 | 71 | 73 | 76 | 78 | 81 | 84 | 87 | 91 | 96 | 101 | 108 | 117 |
| 0.75 | 49 | 53 | 59 | 60 | 62 | 63 | 65 | 67 | 69 | 71 | 73 | 75 | 78 | 81 | 85 | 89 | 94 | 101 | 109 |
| 0.8 | 46 | 50 | 55 | 57 | 58 | 59 | 61 | 63 | 64 | 66 | 68 | 71 | 73 | 76 | 80 | 84 | 89 | 95 | 102 |
| 0.85 | 43 | 47 | 52 | 53 | 55 | 56 | 57 | 59 | 61 | 62 | 64 | 67 | 69 | 72 | 75 | 79 | 83 | 89 | 96 |
| 0.9 | 41 | 44 | 49 | 50 | 52 | 53 | 54 | 56 | 57 | 59 | 61 | 63 | 65 | 68 | 71 | 74 | 79 | 84 | 91 |
| 0.95 | 39 | 42 | 47 | 48 | 49 | 50 | 51 | 53 | 54 | 56 | 58 | 60 | 62 | 64 | 67 | 71 | 75 | 80 | 86 |
| 1 | 37 | 40 | 44 | 45 | 46 | 47 | 49 | 50 | 51 | 53 | 55 | 57 | 59 | 61 | 64 | 67 | 71 | 76 | 82 |

Adapted from Fowler et al., 2019

## **Appendix 2.** Schedule of Events

| | Screen | If Eligible,<br>Baseline<br>Assessment | R | 0<br>hour | 24 (±2)<br>hours | 48 (±2)<br>hours | 72 (±2)<br>hours | 96 (±2)<br>hours | 120 (±2)<br>hours | 144 (±2)<br>hours | 168 hours<br>-Discharge <sup>e</sup> | Day<br>30 <sup>f</sup> | Day<br>60 <sup>f</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Informed Consent | X | | | | | | | | | | | | |
| Weight and Height | X | | | | | | | | | | | | |
| Vital Signs <sup>a</sup> | X | | | | X | X | X | X | X | X | | | |
| P/F ratio | X | | | | X | X | X | X | X | X | | | |
| QTcF | X | | | | X | X | X | X | X | X | | | |
| SARS-CoV-2 testing | X | | | | | | | | | | | | |
| Serum Pregnancy Test in WOCBP | X | | | | | | | | | | | | |
| Daily Laboratory Monitoring | | X | | | X | X | X | X | X | X | | | |
| Nasopharyngeal PCRh | | X | | | | | X <sup>Cohort 1,3</sup> | X <sup>Cohort 2,3</sup> | | | | | |
| $\mathrm{BAL}^{\mathrm{g}}$ | | X | | | | | X <sup>Cohort 1,3</sup> | X <sup>Cohort 2,3</sup> | | | | | |
| Blood for biomarkers | | X | | | | | X <sup>Cohort 1,3</sup> | X <sup>Cohort 2,3</sup> | | | | | |
| PK Analysis | | | | Xb | Xc | Xc | Xc | X <sup>d</sup> | | X | | | |
| AE/SAE/Mortality Assessment | | | | | X | X | X | X | X | X | X | X | X |
| Concomitant Medications | | | | X | X | X | X | X | X | X | | | |
| Randomize patient | | | X | | | | | | | | | | |
| Study Drug Administration | | | | X <sup>Cohorts 1,2,3</sup> | X <sup>Cohorts 1,2</sup> | X <sup>Cohorts 1,2</sup> | X <sup>Cohort 2</sup> | | | | | | |
| Study Drug Continuous Infusion <sup>i</sup> | | | | X <sup>Cohort 3</sup> | X <sup>Cohort 3</sup> | X <sup>Cohort 3</sup> | X <sup>Cohort 3</sup> | | | | | | |

Hospitalized patients will complete all assessments. All patients will complete the Day 30 and Day 60 assessment.

- a. Vital Signs will include temperature, heart rate, respiratory rate, systolic blood pressure, and diastolic blood pressure.
- b. Draw blood sample for PK after finishing the infusion of Auxora (+30 minutes).
- c. For Cohorts 1 and 2 draw blood sample for PK prior to the infusion of Auxora (-2 hours). For Cohort 3, draw PK every 24 hours from SFISD up to hour 72
- d. Draw PK at the end of the continuous infusion (+30 minutes)
- e. In patients who remain hospitalized, AE/SAE/Mortality assessments will be made every 48 hours starting at 168 hours and until Discharge or Day 30, whichever comes first. If patients have been discharged, no follow up during this period is needed; ongoing SAEs should be followed reviewed at Day 30 and Day 60.
- f. Day 30 will be a phone call assessment for patients discharged prior to Day 25. Patients discharged at Days 25,26,27,28,29 will perform the Day 30 assessment before leaving the hospital. Day 60 will be a phone call assessment for patients discharged prior to Day 55 and an inpatient assessment for patients hospitalized between Days 55 and 60.
- g. BAL fluid will be used for flow cytometry, single cell RNA sequencing, and chemokine/biomarker panel. On the post infusion BAL fluid, CM4620 levels will be determined.
- h. Nasopharyngeal swabs will be performed weekly until SARS-CoV-2 RNA is no longer detected
- i. Continuous infusion starts at the end of the first infusion and continues for 96 hours. Infusion ends 100 hours after SFISD